CLINICAL TRIAL: NCT03029247
Title: A Randomized, Open-label Study to Evaluate the Effect of Daprodustat on Blood Pressure in Subjects With Anemia Associated With Chronic Kidney Disease on Hemodialysis Switched From a Stable Dose of an Erythropoiesis-stimulating Agent
Brief Title: Anemia Study in Chronic Kidney Disease (CKD): Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor (PHI) Daprodustat-Blood Pressure (ASCEND-BP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: ERT: Clinical Trial Technology Solutions (Other); Q2 Solutions (Industry); Quintiles, Inc. (Industry); HemoCue (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205665
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Anaemia
Keywords: Anemia; Daprodustat; Blood pressure; ESA; CKD
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants receiving Epoetin alfa (Active Comparator): On Day 1, participants will undergo 24-hour Acute Challenge 1, in which participants will receive a single dose of 100 U/kg epoetin alfa IV. After completing Acute Challenge 1, participants will enter in an 8-week Hgb maintenance period. At the end of Hgb maintenance period, on Day 57, Acute Challenge 2 will be performed utilizing the same treatment dose administered in Acute Challenge 1.
  Interventions: Drug: Epoetin alfa
- Participants receiving Daprodustat (Experimental): On Day 1, participants will undergo 24-hour Acute Challenge 1, in which participants will receive 24 mg daprodustat. After completing Acute Challenge 1, participants will enter an 8-week Hgb maintenance period. At the end of Hgb maintenance period, on Day 57, Acute Challenge 2 will be performed utilizing the same treatment dose administered in Acute Challenge 1.
  Interventions: Drug: Daprodustat

INTERVENTIONS:
Drug: Daprodustat — Daprodustat will be available as oral tablets at unit dose strength of 1, 2, 4, 6, 8 and 10 mg.
  Arms: Participants receiving Daprodustat
Drug: Epoetin alfa — Epoetin alfa will be administered according to local labelling and clinical practice guidelines to keep Hgb in the target range (10.0-11.0 g/dL)
  Arms: Participants receiving Epoetin alfa

SUMMARY:
This will be an open-label, randomized, parallel-group study in hemodialysis-dependent (HD) participants with anemia associated with chronic kidney disease (CKD), designed to compare the effects of daprodustat to epoetin alfa on blood pressure (BP). Participants will be screened for eligibility within 7 and 30 days prior to erythropoesis-stimulating agent (ESA) washout. Following a 2-week ESA washout period, on Day 1 participants will be randomized 1:1 and stratified by prior ESA dose before they undergo Acute Challenge 1, a single dose challenge to compare the acute effects on BP of the highest planned once-daily maintenance dose of daprodustat (24 milligrams [mg]) to the highest starting dose of epoetin alfa (100 units/kilogram [U/kg]). This will be followed by an 8-week hemoglobin (Hgb)-maintenance period, where doses of either daprodustat or epoetin alfa will be administered and adjusted. At the end of Hgb maintenance period, on Day 57 an Acute Challenge 2 will be repeated utilizing the same treatment dose administered in Acute Challenge 1; there will be a follow-up visit within 14+/-3 days after completing treatment.

ELIGIBILITY:
Inclusion Criteria

* More than or equal to 40 years of age, at the time of signing the informed consent
* Stable Hgb 8.5 to 11.5 grams per deciliter (g/dL) inclusive.
* Dialysis frequency: On hemodialysis (HD, hemofiltration or hemodiafiltration) three-to five-times weekly for at least 4 weeks prior to screening.
* A single pool Kt/Vurea >=1.2 based on a historical value obtained within 3 months prior to screening in order to ensure the adequacy of dialysis. If Kt/Vurea is not available, then an average of the last 2 values of urea reduction ratio should be at least 65 percent (%).
* Treated with an ESA (epoetins or their biosimilars, darbepoetin, or methoxy polyethylene glycol [PEG]-epoetin beta) for at least 4 weeks prior to screening.
* Participants may be on stable (<=50% change in overall dose and compliance of 80% of prescribed doses in the 4 weeks prior to and including the screening period) maintenance oral or intravenous (IV; <=100 mg/week) iron supplementation. If participants are on oral or IV iron, then doses must be stable for the 4 weeks prior to Washout.
* Weight: Mid-week weight change between dialysis treatments <5% as assessed post-dialysis at the Screening and Washout visits.
* On at least 1 antihypertensive medication (excluding diuretics) and on that same medication and the same dose for at least 1 week prior to Washout.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and the protocol.
* Willing and able to wear ABPM device for at least 25 hours on two separate sessions.

Exclusion Criteria

* Planned change from HD to peritoneal dialysis within the study time period, or on home dialysis.
* Planned for kidney transplant within the 16 weeks following the Screening visit.
* An epoetin alfa dose of >=360 U/kg/week IV or >=250 U/kg/week subcutaneous (SC), or darbepoetin dose of >=1.8 micrograms (μg)/kg/week IV or SC, or methoxy PEG-epoetin beta dose of >=2.2 μg/kg/week within the 8 weeks prior to screening through Week -4.
* Planned or recorded administration of Mircera (methoxy PEG-epoetin beta) within the 4 weeks prior to the Washout.
* Occurrence of myocardial infarction or acute coronary syndrome within 3 months prior to Washout.
* Stroke or transient ischemic attack within 3 months prior to Washout.
* Chronic Class 4 heart failure, as defined by the New York Heart Association functional classification system diagnosed prior to Washout.
* QT interval corrected for heart rate using Bazett's formula (QTcB) >500 milliseconds (msec), or QTcB >530 msec in participants with Bundle Branch Block. There is no QTc exclusion for participants with a predominantly paced rhythm.
* Resting post dialysis SBP >160 millimeters of mercury (mmHg); or DBP >100 mmHg at screening or uncontrolled hypertension as determined by the investigator.
* Presence of atrial fibrillation.
* Active chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosus, rheumatoid arthritis, celiac disease) diagnosed prior to Washout.
* History of bone marrow aplasia or pure red cell aplasia.
* Other causes of anemia including Pernicious anemia, thalassemia major, sickle cell disease or myelodysplastic syndrome.
* Alanine transaminase (ALT) >2 times upper limit of normal (ULN) (screening only) or Bilirubin >1.5 times ULN (screening only) or Current unstable liver or biliary disease per investigator assessment, generally defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Major surgery (excluding vascular access surgery) within the 3 months prior to Washout or planned during the study.
* Blood transfusion within the 8 weeks prior to Washout or an anticipated need for blood transfusion during the study.
* Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant gastrointestinal bleeding within the 8 weeks prior to Washout.
* Clinical evidence of acute infection or history of infection requiring IV antibiotic therapy within the 8 weeks prior to Washout.
* History of malignancy within the two years prior to screening through Day 1 or currently receiving treatment for cancer, or has a known complex kidney cyst (e.g., Bosniak Category IIF, III or IV) >=3 centimeters.
* Participants with an upper arm diameter which cannot be measured by oscillometer/ sphygmomanometer cuff or for whom BP cannot be measured in the opposite arm of current vascular access.
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product.
* Use of any prescription or non-prescription drugs or dietary supplements that are prohibited from screening until Washout.
* The participant has participated in a clinical trial and has received an experimental investigational product within the 30 days prior to Day 1 or within 5 half lives of the investigational product prior to screening, whichever is longer.
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the participant at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.
* A female participant is pregnant (as confirmed by a positive serum human chorionic gonadotrophin test for females of reproductive potential only), participant is breastfeeding, or participant is of reproductive potential and does not agree to follow one of the pre-specified contraceptive options
* Vitamin B12 at or below the lower limit of the reference range (may rescreen in a minimum of 8 weeks, following treatment).
* Folate at <2.0 nanograms/milliliter (ng/mL) (4.5 Nanomoles per Liter) (may rescreen in a minimum of 4 weeks, following treatment).
* Ferritin at <100 ng/mL
* Transferrin saturation at <20%.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, open label study that evaluated the effect of daprodustat on blood pressure in participants with anemia associated with chronic kidney disease on hemodialysis switched from a stable dose of an erythropoiesis-stimulating agent.
Pre-assignment Details: A total of 105 participants were enrolled of which 88 were randomized to receive study treatment. 17 did not receive study treatment as they were withdrawn prior to randomization due to adverse events (2); protocol deviation (2); protocol specified withdrawal criteria (3); lost to follow-up (1); physician decision (2) and withdrawal by participant (7).
Groups:
- Daprodustat: Participants were randomized to receive a single oral dose of Daprodustat 24 milligrams (mg) during 24-hour acute challenge 1 (AC1) on Day 1. Participants discontinued their current erythropoiesis stimulating agent (ESA) therapy and were washed out of their ESAs for 2 weeks prior to acute challenge 1. After completion of acute challenge 1, participants entered in 8-week hemoglobin (Hgb) maintenance period, where doses of daprodustat were administered and adjusted to maintain target Hgb levels within the range of 10.0 to 11.0 grams per deciliter (g/dL). Participants received acute challenge 2 (AC2) on Day 57 with the same treatment dose administered in acute challenge 1. All participants were followed up for 14 days after acute challenge 2.
- Recombinant Human Erythropoietin: Participants were randomized to receive a single intravenous (IV) dose of 100 units per kilogram (U/Kg) Epoetin alfa (Recombinant human erythropoietin) during 24-hour acute challenge 1 on Day 1. Participants discontinued their current ESA therapy and were washed out of their ESAs for 2 weeks prior to acute challenge 1. After completion of acute challenge 1, participants entered in 8-week Hgb maintenance period, where Epoetin alfa was administered according to local labelling and clinical practice guidelines to maintain target Hgb levels within the range of 10.0 to 11.0 g/dL. Participants received acute challenge 2 on Day 57 with the same treatment dose administered in acute challenge 1. All participants were followed up for 14 days after acute challenge 2.
Period: Acute Challenge 1 (Day 1)
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Started | 45 | 43
Completed | 45 | 43
Not Completed | 0 | 0
Period: Hgb Maintenance Phase (8 Weeks)
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Started | 45 | 43
Completed | 32 | 36
Not Completed | 13 | 7
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol-specified withdrawal criterion | 7 | 4
Not completed — Adverse Event | 2 | 2
Period: Acute Challenge 2 (Day 57)
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Started | 32 | 36
Completed | 32 | 36
Not Completed | 0 | 0
Period: Follow-up Period (14 Days)
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Started | 32 | 36
Completed | 32 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | Recombinant Human Erythropoietin | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (11.06) | 58.7 (10.61) | 59.8 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 26 | 27 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 21 | 23 | 44
  White-Arabic/North African Heritage | 1 | 0 | 1
  White-White/Caucasian/European Heritage | 23 | 20 | 43

OUTCOME MEASURES:

1. Primary Outcome: Average of Systolic Blood Pressure (SBP) Measured by Ambulatory Blood Pressure Monitoring (ABPM) Over 6-hour Post Dosing on Day 57
Description: The effect of daprodustat and epoetin alfa on blood pressure was compared using ABPM after 8 weeks of Hgb maintenace therapy on Day 57. Analysis was based on "analysis of covariance (ANCOVA) with terms for treatment, prior erythropoiesis-stimulating agent (ESA) dose (low/high), post-Hemodialysis dependent (HD)/pre-AC 1 SBP, difference between post-HD/pre-AC 2 SBP and post-HD/pre-AC 1 SBP and treatment by difference in post-HD SBP between AC 1 and 2 interaction." Least square (LS) mean of 6 hour average SBP post AC2 on Day 57 and its corresponding standard error has been presented.
Time Frame: Up to 6 hours post dose on Day 57
Population: Intent-to-Treat (ITT)-Population comprised of all randomized participants who received at least one dose of study treatment. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeters of mercury (mmHg)
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 27 | 28
Millimeters of mercury (mmHg) | 142.87 (3.039) | 143.03 (2.995)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.9694, ANCOVA — p-value for the difference between treatment groups were presented from ANCOVA model for the superiority assessment; LS Mean Difference = -0.17, 95% CI 2-sided [-8.80 to 8.47] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) and its corresponding 95% confidence interval (CI) has been presented

2. Secondary Outcome: Average of SBP, Diastolic Blood Pressure (DBP) and Mean Arterial Blood Pressure (MAP) Measured by ABPM Over 6-hour Post Dosing on Day 1
Description: The initial effect of daprodustat and epoetin alfa on blood pressure was compared using ABPM over 6 hour post-dosing on Day 1. Analysis was based on ANCOVA with terms for treatment, prior ESA dose (low/high), post-HD/pre-AC1 SBP, DBP and MAP. LS mean of 6 hour average SBP, DBP and MAP post AC1 on Day 1 and its corresponding standard error has been presented.
Time Frame: Up to 6 hours post dose on Day 1
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 35 | 31
mmHg
  SBP | 141.36 (3.115) | 142.68 (3.313)
  DBP | 75.97 (1.253) | 77.92 (1.332)
  MAP | 99.18 (2.212) | 101.58 (2.351)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.7745, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -1.32, 95% CI 2-sided [-10.46 to 7.83] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) of SBP and its corresponding 95% CI has been presented
Statistical Analysis 2: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.2910, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -1.95, 95% CI 2-sided [-5.62 to 1.71] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) of DBP and its corresponding 95% CI has been presented
Statistical Analysis 3: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.4611, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -2.40, 95% CI 2-sided [-8.88 to 4.07] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) of MAP and its corresponding 95% CI has been presented

3. Secondary Outcome: Average of Heart Rate (HR) Measured by ABPM Over 6 Hour Post Dosing on Day 1
Description: The initial effect of daprodustat and epoetin alfa on HR was compared using ABPM over 6 hour post-dosing on Day 1. Analysis was based on ANCOVA with terms for treatment, prior ESA dose (low/high), post-HD/pre-AC1 HR. LS mean of 6 hour average HR post AC1 on Day 1 and its corresponding standard error has been presented.
Time Frame: Up to 6 hours post dose on Day 1
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 35 | 31
Beats per minute | 70.77 (1.416) | 73.72 (1.507)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.1648, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -2.95, 95% CI 2-sided [-7.14 to 1.24] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) and its corresponding 95% CI has been presented

4. Secondary Outcome: Area Under the Effect Curve (AUEC) of SBP, DBP and MAP Measured by ABPM Over 24-hour Post Dosing on Day 1
Description: The initial effect of daprodustat and epoetin alfa on blood pressure was compared using AUEC of SBP, DBP and MAP measured by ABPM over 24-hour post dosing on Day 1. Analysis was based on ANCOVA with terms for treatment and prior ESA dose (low/high). LS mean of AUEC up to 24 hours post dose on Day 1 and its corresponding standard error has been presented.
Time Frame: Up to 24 hours post dose on Day 1
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg*Hours
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 31 | 27
mmHg*Hours
  AUEC of SBP | 3337.91 (84.144) | 3351.33 (90.217)
  AUEC of DBP | 1763.11 (39.814) | 1834.82 (42.688)
  AUEC of MAP | 2324.69 (57.517) | 2378.93 (61.668)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.9142, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -13.42, 95% CI 2-sided [-261.75 to 234.92] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) for AUEC of SBP and its corresponding 95% CI has been presented
Statistical Analysis 2: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.2266, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -71.70, 95% CI 2-sided [-189.21 to 45.80] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) for AUEC of DBP and its corresponding 95% CI has been presented
Statistical Analysis 3: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.5246, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -54.24, 95% CI 2-sided [-223.99 to 115.51] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) for AUEC of MAP and its corresponding 95% CI has been presented

5. Secondary Outcome: AUEC of HR Measured by ABPM Over 24-hour Post Dosing on Day 1
Description: The initial effect of daprodustat and epoetin alfa on HR was compared using AUEC of HR measured by ABPM over 24-hour post dosing. Analysis was based on ANCOVA with terms for treatment and prior ESA dose (low/high). LS mean of AUEC up to 24 hours post dose on Day 1 and its corresponding standard error has been presented.
Time Frame: Up to 24 hours post dose on Day 1
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute*Hours
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 31 | 27
Beats per minute*Hours | 1652.63 (35.152) | 1727.03 (37.690)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.1563, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -74.40, 95% CI 2-sided [-178.15 to 29.34] — LS Mean treatment difference (daprodustat minus recombinant human erythropoietin) for AUEC of HR and its corresponding 95% CI has been presented

6. Secondary Outcome: Average of DBP and MAP Measured by ABPM Over 6-hour Post Dosing on Day 57
Description: The effect of daprodustat and epoetin alfa on blood pressure was compared using ABPM over 6 hour post-dosing after AC2 on Day 57. Analysis was based on ANCOVA with terms for treatment, prior ESA dose (low/high), post-HD/pre-AC1 DBP and MAP, difference between post-HD/pre-AC2 DBP and MAP and post-HD/pre-AC1 DBP and MAP and treatment by difference in post-HD DBP and MAP between AC1 and 2 interaction. LS mean of 6 hour average DBP and MAP post AC2 on Day 57 and its corresponding standard error has been presented.
Time Frame: Up to 6 hours post dose on Day 57
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 27 | 28
mmHg
  DBP | 75.58 (1.465) | 77.64 (1.436)
  MAP | 98.98 (2.208) | 101.49 (2.169)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.3247, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -2.06, 95% CI 2-sided [-6.23 to 2.10] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.4235, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -2.51, 95% CI 2-sided [-8.76 to 3.74] — [estimate comment as in outcome 2, analysis 3]

7. Secondary Outcome: Average of HR Measured by ABPM Over 6 Hour Post Dosing on Day 57
Description: The effect of daprodustat and epoetin alfa on HR was compared using ABPM over 6 hour post-dosing. Analysis was based on ANCOVA with terms for treatment, prior ESA dose (low/high), post-HD/pre-AC1 HR, difference between post-HD/pre-AC2 HR and post-HD/pre-AC1 HR and treatment by difference in post-HD HR between AC1 and 2 interaction. LS mean of 6 hour average HR post AC2 on Day 57 and its corresponding standard error has been presented.
Time Frame: Up to 6 hours post dose on Day 57
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 27 | 28
Beats per minute | 70.49 (1.146) | 70.62 (1.125)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.9353, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -0.13, 95% CI 2-sided [-3.41 to 3.14] — [estimate comment as in outcome 3, analysis 1]

8. Secondary Outcome: AUEC of SBP, DBP and MAP Measured by ABPM Over 24-hour Post Dosing on Day 57
Description: The effect of daprodustat and epoetin alfa on blood pressure was compared using AUEC of SBP, DBP and MAP measured by ABPM over 24-hour post dosing on Day 57. Analysis was based on ANCOVA with terms for treatment and prior ESA dose (low/high). LS mean of AUEC up to 24 hour post dose on Day 57 and its corresponding standard error has been presented.
Time Frame: Up to 24 hours post dose on Day 57
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mmHg*Hours
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 24 | 21
mmHg*Hours
  AUEC of SBP | 3288.43 (85.805) | 3433.40 (91.786)
  AUEC of DBP | 1736.11 (38.659) | 1853.60 (41.354)
  AUEC of MAP | 2299.42 (58.712) | 2431.36 (62.804)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.2573, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -144.97, 95% CI 2-sided [-399.71 to 109.76] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.0450, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -117.49, 95% CI 2-sided [-232.26 to -2.72] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.1341, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -131.94, 95% CI 2-sided [-306.24 to 42.36] — [estimate comment as in outcome 4, analysis 3]

9. Secondary Outcome: AUEC of HR Measured by ABPM Over 24-hour Post Dosing on Day 57
Description: The effect of daprodustat and epoetin alfa on HR was compared using AUEC of HR measured by ABPM over 24-hour post dosing on Day 57. Analysis was based on ANCOVA with terms for treatment and prior ESA dose (low/high). LS mean of AUEC up to 24 hour post dose on Day 57 and its corresponding standard error has been presented.
Time Frame: Up to 24 hours post dose on Day 57
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Beats per minute*Hours
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 24 | 21
Beats per minute*Hours | 1579.38 (40.886) | 1677.06 (43.736)
Statistical Analysis 1: Comparison: Daprodustat vs Recombinant Human Erythropoietin; Test type: Superiority; p = 0.1119, ANCOVA — p-value for the difference between treatment groups was presented from ANCOVA model for the superiority assessment; LS Mean Difference = -97.67, 95% CI 2-sided [-219.05 to 23.71] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Change From Pre-dose in SBP, DBP and MAP at Day 1
Description: The change from pre-dose in SBP, DBP and MAP was measured using ABPM to compare the initial effect of daprodustat to epoetin alfa after AC1 on Day 1. Change from pre-dose at each timepoint is calculated as measurement at post-dose minus pre-acute challenge 1 measurement.
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23 and 24 hours post-dose
Population: ITT-Population. Only those participants with data available at specified time points has been presented (represented as n=X in category titles).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 35 | 31
mmHg
  SBP, Hour 1, n=34, 31: number analyzed (Participants) | 34 | 31
  SBP, Hour 1, n=34, 31 | 1.00 (17.178) | 5.27 (20.471)
  SBP, Hour 2, n=35, 31 | -4.99 (28.170) | 4.72 (22.651)
  SBP, Hour 3, n=35, 31 | -5.85 (29.636) | 5.09 (21.163)
  SBP, Hour 4, n=35, 31 | -1.68 (26.000) | 0.93 (23.962)
  SBP, Hour 5, n=35, 31 | -1.86 (29.171) | -2.10 (23.849)
  SBP, Hour 6, n=35, 31 | 0.29 (31.903) | -2.54 (28.908)
  SBP, Hour 7, n=34, 26: number analyzed (Participants) | 34 | 26
  SBP, Hour 7, n=34, 26 | 2.30 (33.896) | 0.63 (19.016)
  SBP, Hour 8, n=33, 29: number analyzed (Participants) | 33 | 29
  SBP, Hour 8, n=33, 29 | 0.43 (31.418) | 3.83 (20.723)
  SBP, Hour 9, n=33, 30: number analyzed (Participants) | 33 | 30
  SBP, Hour 9, n=33, 30 | -5.81 (30.725) | 0.25 (26.294)
  SBP, Hour 10, n=31, 28: number analyzed (Participants) | 31 | 28
  SBP, Hour 10, n=31, 28 | -5.70 (28.018) | 1.48 (25.952)
  SBP, Hour 11, n=33, 27: number analyzed (Participants) | 33 | 27
  SBP, Hour 11, n=33, 27 | -7.00 (27.529) | 1.96 (24.421)
  SBP, Hour 12, n=35, 28: number analyzed (Participants) | 35 | 28
  SBP, Hour 12, n=35, 28 | -6.05 (29.932) | -1.67 (19.380)
  SBP, Hour 13, n=34, 28: number analyzed (Participants) | 34 | 28
  SBP, Hour 13, n=34, 28 | -2.49 (25.319) | -1.37 (25.596)
  SBP, Hour 14, n=34, 31: number analyzed (Participants) | 34 | 31
  SBP, Hour 14, n=34, 31 | -5.30 (30.030) | 4.57 (29.767)
  SBP, Hour 15, n=32, 26: number analyzed (Participants) | 32 | 26
  SBP, Hour 15, n=32, 26 | -1.47 (33.573) | -0.13 (24.287)
  SBP, Hour 16, n=34, 31: number analyzed (Participants) | 34 | 31
  SBP, Hour 16, n=34, 31 | -4.40 (30.990) | 8.59 (24.729)
  SBP, Hour 17, n=32, 30: number analyzed (Participants) | 32 | 30
  SBP, Hour 17, n=32, 30 | -5.05 (29.795) | 1.76 (23.896)
  SBP, Hour 18, n=32, 27: number analyzed (Participants) | 32 | 27
  SBP, Hour 18, n=32, 27 | -5.23 (25.993) | 5.48 (23.330)
  SBP, Hour 19, n=34, 27: number analyzed (Participants) | 34 | 27
  SBP, Hour 19, n=34, 27 | -3.01 (24.230) | 1.52 (21.072)
  SBP, Hour 20, n=33, 27: number analyzed (Participants) | 33 | 27
  SBP, Hour 20, n=33, 27 | -13.27 (24.138) | 6.89 (16.834)
  SBP, Hour 21, n=30, 27: number analyzed (Participants) | 30 | 27
  SBP, Hour 21, n=30, 27 | -8.32 (26.003) | 1.72 (26.777)
  SBP, Hour 22, n=29, 27: number analyzed (Participants) | 29 | 27
  SBP, Hour 22, n=29, 27 | -3.93 (26.106) | 3.50 (24.428)
  SBP, Hour 23, n=31, 26: number analyzed (Participants) | 31 | 26
  SBP, Hour 23, n=31, 26 | 2.73 (28.343) | 8.72 (24.868)
  SBP, Hour 24, n=31, 27: number analyzed (Participants) | 31 | 27
  SBP, Hour 24, n=31, 27 | 2.63 (29.379) | 5.02 (26.601)
  DBP, Hour 1, n=34, 31: number analyzed (Participants) | 34 | 31
  DBP, Hour 1, n=34, 31 | 0.01 (9.317) | 0.99 (13.110)
  DBP, Hour 2, n=35, 31 | -0.82 (15.399) | 1.97 (11.986)
  DBP, Hour 3, n=35, 31 | -1.30 (14.660) | 0.88 (11.858)
  DBP, Hour 4, n=35, 31 | -1.06 (14.552) | -1.17 (13.621)
  DBP, Hour 5, n=35, 31 | -0.69 (16.618) | -1.49 (11.684)
  DBP, Hour 6, n=35, 31 | -0.06 (14.799) | -1.49 (14.457)
  DBP, Hour 7, n=34, 26: number analyzed (Participants) | 34 | 26
  DBP, Hour 7, n=34, 26 | -0.12 (16.324) | -1.27 (15.272)
  DBP, Hour 8, n=33, 29: number analyzed (Participants) | 33 | 29
  DBP, Hour 8, n=33, 29 | 1.35 (15.900) | 1.79 (15.178)
  DBP, Hour 9, n=33, 30: number analyzed (Participants) | 33 | 30
  DBP, Hour 9, n=33, 30 | -2.14 (15.188) | -0.68 (11.874)
  DBP, Hour 10, n=31, 28: number analyzed (Participants) | 31 | 28
  DBP, Hour 10, n=31, 28 | -3.52 (14.246) | -0.82 (12.802)
  DBP, Hour 11, n=33, 27: number analyzed (Participants) | 33 | 27
  DBP, Hour 11, n=33, 27 | -4.88 (14.691) | -2.45 (10.987)
  DBP, Hour 12, n=35, 28: number analyzed (Participants) | 35 | 28
  DBP, Hour 12, n=35, 28 | -4.79 (14.561) | -3.95 (10.718)
  DBP, Hour 13, n=34, 28: number analyzed (Participants) | 34 | 28
  DBP, Hour 13, n=34, 28 | -2.15 (15.185) | -2.65 (12.841)
  DBP, Hour 14, n=34, 31: number analyzed (Participants) | 34 | 31
  DBP, Hour 14, n=34, 31 | -3.99 (14.153) | -1.00 (14.759)
  DBP, Hour 15, n=32, 26: number analyzed (Participants) | 32 | 26
  DBP, Hour 15, n=32, 26 | -0.54 (19.203) | -4.12 (13.905)
  DBP, Hour 16, n=34, 31: number analyzed (Participants) | 34 | 31
  DBP, Hour 16, n=34, 31 | -3.56 (15.615) | 1.15 (14.186)
  DBP, Hour 17, n=32, 30: number analyzed (Participants) | 32 | 30
  DBP, Hour 17, n=32, 30 | -3.65 (14.949) | -2.98 (13.732)
  DBP, Hour 18, n=32, 27: number analyzed (Participants) | 32 | 27
  DBP, Hour 18, n=32, 27 | -2.08 (17.015) | 0.30 (14.219)
  DBP, Hour 19, n=34, 27: number analyzed (Participants) | 34 | 27
  DBP, Hour 19, n=34, 27 | -0.36 (19.650) | -0.43 (14.965)
  DBP, Hour 20, n=33, 27: number analyzed (Participants) | 33 | 27
  DBP, Hour 20, n=33, 27 | -2.96 (15.579) | 0.40 (14.501)
  DBP, Hour 21, n=30, 27: number analyzed (Participants) | 30 | 27
  DBP, Hour 21, n=30, 27 | -2.54 (15.246) | 1.90 (15.507)
  DBP, Hour 22, n=29, 27: number analyzed (Participants) | 29 | 27
  DBP, Hour 22, n=29, 27 | -0.25 (15.037) | -1.96 (12.058)
  DBP, Hour 23, n=31, 26: number analyzed (Participants) | 31 | 26
  DBP, Hour 23, n=31, 26 | 4.05 (19.055) | -0.44 (13.218)
  DBP, Hour 24, n=31, 27: number analyzed (Participants) | 31 | 27
  DBP, Hour 24, n=31, 27 | 4.48 (18.097) | 2.16 (15.124)
  MAP, Hour 1, n=34, 31: number analyzed (Participants) | 34 | 31
  MAP, Hour 1, n=34, 31 | -1.87 (15.252) | 2.83 (19.439)
  MAP, Hour 2, n=35, 31 | -4.79 (24.742) | 4.20 (17.890)
  MAP, Hour 3, n=35, 31 | -5.13 (22.342) | 3.46 (14.940)
  MAP, Hour 4, n=35, 31 | -4.78 (23.640) | -1.05 (17.552)
  MAP, Hour 5, n=35, 31 | -3.48 (26.458) | -1.18 (16.235)
  MAP, Hour 6, n=35, 31 | -1.27 (25.359) | -2.17 (19.573)
  MAP, Hour 7, n=34, 26: number analyzed (Participants) | 34 | 26
  MAP, Hour 7, n=34, 26 | 0.45 (28.445) | 0.87 (18.659)
  MAP, Hour 8, n=33, 29: number analyzed (Participants) | 33 | 29
  MAP, Hour 8, n=33, 29 | 0.08 (27.487) | 2.20 (17.002)
  MAP, Hour 9, n=33, 30: number analyzed (Participants) | 33 | 30
  MAP, Hour 9, n=33, 30 | -7.02 (24.498) | 0.61 (17.072)
  MAP, Hour 10, n=31, 28: number analyzed (Participants) | 31 | 28
  MAP, Hour 10, n=31, 28 | -8.18 (24.057) | 0.76 (18.604)
  MAP, Hour 11, n=33, 27: number analyzed (Participants) | 33 | 27
  MAP, Hour 11, n=33, 27 | -8.74 (25.719) | -3.60 (19.022)
  MAP, Hour 12, n=35, 28: number analyzed (Participants) | 35 | 28
  MAP, Hour 12, n=35, 28 | -6.49 (26.669) | -6.15 (16.336)
  MAP, Hour 13, n=34, 28: number analyzed (Participants) | 34 | 28
  MAP, Hour 13, n=34, 28 | -5.72 (23.609) | -3.32 (17.660)
  MAP, Hour 14, n=34, 31: number analyzed (Participants) | 34 | 31
  MAP, Hour 14, n=34, 31 | -6.99 (25.710) | -0.75 (17.024)
  MAP, Hour 15, n=32, 26: number analyzed (Participants) | 32 | 26
  MAP, Hour 15, n=32, 26 | -4.06 (27.693) | -5.10 (19.458)
  MAP, Hour 16, n=34, 31: number analyzed (Participants) | 34 | 31
  MAP, Hour 16, n=34, 31 | -4.79 (26.805) | 3.84 (22.886)
  MAP, Hour 17, n=32, 30: number analyzed (Participants) | 32 | 30
  MAP, Hour 17, n=32, 30 | -5.10 (25.873) | -2.09 (19.856)
  MAP, Hour 18, n=32, 27: number analyzed (Participants) | 32 | 27
  MAP, Hour 18, n=32, 27 | -6.98 (24.790) | 1.52 (18.745)
  MAP, Hour 19, n=34, 27: number analyzed (Participants) | 34 | 27
  MAP, Hour 19, n=34, 27 | -4.44 (26.186) | -1.02 (17.275)
  MAP, Hour 20, n=33, 27: number analyzed (Participants) | 33 | 27
  MAP, Hour 20, n=33, 27 | -9.47 (23.186) | 4.23 (16.311)
  MAP, Hour 21, n=30, 27: number analyzed (Participants) | 30 | 27
  MAP, Hour 21, n=30, 27 | -7.39 (22.611) | 3.87 (20.860)
  MAP, Hour 22, n=29, 27: number analyzed (Participants) | 29 | 27
  MAP, Hour 22, n=29, 27 | -2.77 (21.938) | 0.75 (16.888)
  MAP, Hour 23, n=31, 26: number analyzed (Participants) | 31 | 26
  MAP, Hour 23, n=31, 26 | 0.88 (27.381) | 4.10 (18.818)
  MAP, Hour 24, n=31, 27: number analyzed (Participants) | 31 | 27
  MAP, Hour 24, n=31, 27 | 2.02 (26.253) | 2.20 (19.276)

11. Secondary Outcome: Change From Pre-dose in HR at Day 1
Description: The change from pre-dose in HR was measured using ABPM to compare the initial effect of daprodustat to epoetin alfa after AC1 on Day 1. Change from pre-dose at each timepoint is calculated as measurement at post-dose minus pre-acute challenge 1 measurement.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 35 | 31
Beats per minute
  Hour 1, n=34, 31: number analyzed (Participants) | 34 | 31
  Hour 1, n=34, 31 | -1.16 (9.283) | 0.13 (15.465)
  Hour 2, n=35, 31 | -1.05 (17.259) | -2.06 (15.409)
  Hour 3, n=35, 31 | 0.76 (15.920) | -0.16 (14.911)
  Hour 4, n=35, 31 | 3.18 (12.717) | -1.13 (17.798)
  Hour 5, n=35, 31 | 0.91 (13.782) | -0.66 (14.119)
  Hour 6, n=35, 31 | 0.97 (14.763) | -1.66 (13.023)
  Hour 7, n=34, 26: number analyzed (Participants) | 34 | 26
  Hour 7, n=34, 26 | 2.14 (13.620) | -1.01 (11.592)
  Hour 8, n=33, 29: number analyzed (Participants) | 33 | 29
  Hour 8, n=33, 29 | 0.62 (13.326) | -1.11 (18.376)
  Hour 9, n=33, 30: number analyzed (Participants) | 33 | 30
  Hour 9, n=33, 30 | 0.20 (14.533) | 0.67 (15.411)
  Hour 10, n=31, 28: number analyzed (Participants) | 31 | 28
  Hour 10, n=31, 28 | 2.54 (13.575) | 1.60 (13.612)
  Hour 11, n=33, 27: number analyzed (Participants) | 33 | 27
  Hour 11, n=33, 27 | 2.07 (14.247) | 1.57 (14.132)
  Hour 12, n=35, 28: number analyzed (Participants) | 35 | 28
  Hour 12, n=35, 28 | 0.77 (12.386) | -2.01 (14.767)
  Hour 13, n=34, 28: number analyzed (Participants) | 34 | 28
  Hour 13, n=34, 28 | -0.25 (12.895) | -2.45 (14.861)
  Hour 14, n=34, 31: number analyzed (Participants) | 34 | 31
  Hour 14, n=34, 31 | -1.54 (13.148) | 0.25 (13.020)
  Hour 15, n=32, 26: number analyzed (Participants) | 32 | 26
  Hour 15, n=32, 26 | -0.92 (13.406) | -3.06 (13.156)
  Hour 16, n=34, 31: number analyzed (Participants) | 34 | 31
  Hour 16, n=34, 31 | -1.02 (14.018) | -2.87 (11.762)
  Hour 17, n=32, 30: number analyzed (Participants) | 32 | 30
  Hour 17, n=32, 30 | -0.85 (14.631) | -4.34 (13.284)
  Hour 18, n=32, 27: number analyzed (Participants) | 32 | 27
  Hour 18, n=32, 27 | 0.60 (15.553) | 0.98 (11.443)
  Hour 19, n=34, 27: number analyzed (Participants) | 34 | 27
  Hour 19, n=34, 27 | -0.56 (14.407) | -2.65 (13.220)
  Hour 20, n=33, 27: number analyzed (Participants) | 33 | 27
  Hour 20, n=33, 27 | -1.91 (13.956) | -4.77 (17.083)
  Hour 21, n=30, 27: number analyzed (Participants) | 30 | 27
  Hour 21, n=30, 27 | -1.82 (13.841) | -3.00 (13.342)
  Hour 22, n=29, 27: number analyzed (Participants) | 29 | 27
  Hour 22, n=29, 27 | 0.82 (11.686) | -2.61 (13.292)
  Hour 23, n=31, 26: number analyzed (Participants) | 31 | 26
  Hour 23, n=31, 26 | -1.01 (12.697) | 0.24 (13.148)
  Hour 24, n=31, 27: number analyzed (Participants) | 31 | 27
  Hour 24, n=31, 27 | -0.89 (17.530) | -0.96 (14.651)

12. Secondary Outcome: Plasma Concentrations of Daprodustat
Description: Blood samples were collected at indicated time points for the concentrations of daprodustat.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: Pharmacokinetic Population comprised of all participants in the Safety population who had at least 1 non-missing pharmacokinetic assessment. Only those participants with data available at specified time points has been presented (represented as n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 197.118 (329.0251)
  Day 1, 1 hour, n=43: number analyzed (Participants) | 43
  Day 1, 1 hour, n=43 | 265.828 (340.7690)
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 156.103 (150.4148)
  Day 1, 3 hours, n=43: number analyzed (Participants) | 43
  Day 1, 3 hours, n=43 | 114.485 (139.8114)
  Day 1, 4 hours, n=44: number analyzed (Participants) | 44
  Day 1, 4 hours, n=44 | 105.375 (150.0982)
  Day 1, 6 hours, n=44: number analyzed (Participants) | 44
  Day 1, 6 hours, n=44 | 71.995 (104.2462)
  Day 1, 8 hours, n=43: number analyzed (Participants) | 43
  Day 1, 8 hours, n=43 | 50.069 (91.2574)
  Day 1, 12 hours, n=41: number analyzed (Participants) | 41
  Day 1, 12 hours, n=41 | 14.165 (30.2719)
  Day 1, 16 hours, n=43: number analyzed (Participants) | 43
  Day 1, 16 hours, n=43 | 5.350 (11.0233)
  Day 1, 24 hours, n=43: number analyzed (Participants) | 43
  Day 1, 24 hours, n=43 | 2.899 (10.8052)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 8.657 (21.3825)
  Day 57, 0.5 hours, n=31: number analyzed (Participants) | 31
  Day 57, 0.5 hours, n=31 | 175.616 (257.3578)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 260.817 (307.2242)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 245.277 (251.2676)
  Day 57, 3 hours, n=31: number analyzed (Participants) | 31
  Day 57, 3 hours, n=31 | 142.366 (154.9041)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 82.696 (104.8654)
  Day 57, 6 hours, n=31: number analyzed (Participants) | 31
  Day 57, 6 hours, n=31 | 43.751 (55.8532)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 16.484 (27.2733)
  Day 57, 12 hours, n=30: number analyzed (Participants) | 30
  Day 57, 12 hours, n=30 | 8.661 (16.8915)
  Day 57, 16 hours, n=30: number analyzed (Participants) | 30
  Day 57, 16 hours, n=30 | 7.279 (21.2784)
  Day 57, 24 hours, n=31: number analyzed (Participants) | 31
  Day 57, 24 hours, n=31 | 1.371 (2.0177)

13. Secondary Outcome: Plasma Concentrations of Metabolite GSK2391220
Description: Blood samples were collected at indicated time points for the concentrations of metabolite GSK2391220.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: Pharmacokinetic Population. Only those participants with data available at specified time points has been presented (represented as n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 9.847 (NA) — Not applicable (NA) indicates Standard deviation (SD) could not be calculated due to the high proportion of non-quantifiable (NQ) values (>30% of values were imputed) which affected the SD.
  Day 1, 1 hour, n=43: number analyzed (Participants) | 43
  Day 1, 1 hour, n=43 | 14.361 (21.6405)
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 30.036 (29.6152)
  Day 1, 3 hours, n=44: number analyzed (Participants) | 44
  Day 1, 3 hours, n=44 | 32.359 (28.6734)
  Day 1, 4 hours, n=43: number analyzed (Participants) | 43
  Day 1, 4 hours, n=43 | 32.892 (27.2772)
  Day 1, 6 hours, n=43: number analyzed (Participants) | 43
  Day 1, 6 hours, n=43 | 33.105 (20.9136)
  Day 1, 8 hours, n=42: number analyzed (Participants) | 42
  Day 1, 8 hours, n=42 | 32.267 (16.3824)
  Day 1, 12 hours, n=40: number analyzed (Participants) | 40
  Day 1, 12 hours, n=40 | 23.921 (15.1007)
  Day 1, 16 hours, n=42: number analyzed (Participants) | 42
  Day 1, 16 hours, n=42 | 19.771 (13.5013)
  Day 1, 24 hours, n=42: number analyzed (Participants) | 42
  Day 1, 24 hours, n=42 | 12.693 (10.1135)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 3.019 (4.2327)
  Day 57, 0.5 hours, n=31: number analyzed (Participants) | 31
  Day 57, 0.5 hours, n=31 | 10.043 (12.5832)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 12.410 (13.3576)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 23.433 (21.4154)
  Day 57, 3 hours, n=31: number analyzed (Participants) | 31
  Day 57, 3 hours, n=31 | 32.861 (26.3829)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 38.443 (27.9354)
  Day 57, 6 hours, n=31: number analyzed (Participants) | 31
  Day 57, 6 hours, n=31 | 41.432 (24.2976)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 33.689 (20.3669)
  Day 57, 12 hours, n=31: number analyzed (Participants) | 31
  Day 57, 12 hours, n=31 | 25.771 (17.8554)
  Day 57, 16 hours, n=31: number analyzed (Participants) | 31
  Day 57, 16 hours, n=31 | 21.481 (15.6404)
  Day 57, 24 hours, n=32: number analyzed (Participants) | 32
  Day 57, 24 hours, n=32 | 14.836 (11.2824)

14. Secondary Outcome: Plasma Concentrations of Metabolite GSK2506104
Description: Blood samples were collected at indicated time points for the concentrations of metabolite GSK2506104.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 9.337 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 1 hour, n=43: number analyzed (Participants) | 43
  Day 1, 1 hour, n=43 | 13.263 (20.5510)
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 28.986 (28.4324)
  Day 1, 3 hours, n=44: number analyzed (Participants) | 44
  Day 1, 3 hours, n=44 | 32.623 (29.1622)
  Day 1, 4 hours, n=43: number analyzed (Participants) | 43
  Day 1, 4 hours, n=43 | 34.266 (27.5021)
  Day 1, 6 hours, n=43: number analyzed (Participants) | 43
  Day 1, 6 hours, n=43 | 37.250 (21.9404)
  Day 1, 8 hours, n=42: number analyzed (Participants) | 42
  Day 1, 8 hours, n=42 | 39.463 (17.2013)
  Day 1, 12 hours, n=40: number analyzed (Participants) | 40
  Day 1, 12 hours, n=40 | 33.822 (16.6962)
  Day 1, 16 hours, n=42: number analyzed (Participants) | 42
  Day 1, 16 hours, n=42 | 31.224 (16.3048)
  Day 1, 24 hours, n=42: number analyzed (Participants) | 42
  Day 1, 24 hours, n=42 | 24.268 (14.2298)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 4.133 (4.5315)
  Day 57, 0.5 hours, n=31: number analyzed (Participants) | 31
  Day 57, 0.5 hours, n=31 | 10.759 (11.6369)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 12.902 (12.5068)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 23.391 (20.1627)
  Day 57, 3 hours, n=31: number analyzed (Participants) | 31
  Day 57, 3 hours, n=31 | 33.561 (26.4516)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 41.089 (28.8815)
  Day 57, 6 hours, n=31: number analyzed (Participants) | 31
  Day 57, 6 hours, n=31 | 47.511 (25.5686)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 43.646 (22.0075)
  Day 57, 12 hours, n=31: number analyzed (Participants) | 31
  Day 57, 12 hours, n=31 | 39.685 (23.4732)
  Day 57, 16 hours, n=31: number analyzed (Participants) | 31
  Day 57, 16 hours, n=31 | 36.234 (22.1830)
  Day 57, 24 hours, n=32: number analyzed (Participants) | 32
  Day 57, 24 hours, n=32 | 27.808 (14.8739)

15. Secondary Outcome: Plasma Concentrations of Metabolite GSK2487818
Description: Blood samples were collected at indicated time points for the concentrations of metabolite GSK2487818.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 8.624 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 1 hour, n=43: number analyzed (Participants) | 43
  Day 1, 1 hour, n=43 | 13.181 (19.2280)
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 25.204 (24.8233)
  Day 1, 3 hours, n=44: number analyzed (Participants) | 44
  Day 1, 3 hours, n=44 | 23.632 (21.0661)
  Day 1, 4 hours, n=43: number analyzed (Participants) | 43
  Day 1, 4 hours, n=43 | 20.726 (17.9713)
  Day 1, 6 hours, n=43: number analyzed (Participants) | 43
  Day 1, 6 hours, n=43 | 15.509 (10.4545)
  Day 1, 8 hours, n=42: number analyzed (Participants) | 42
  Day 1, 8 hours, n=42 | 11.654 (9.1747)
  Day 1, 12 hours, n=39: number analyzed (Participants) | 39
  Day 1, 12 hours, n=39 | 5.673 (6.4670)
  Day 1, 16 hours, n=43: number analyzed (Participants) | 43
  Day 1, 16 hours, n=43 | 3.298 (4.6779)
  Day 1, 24 hours, n=43: number analyzed (Participants) | 43
  Day 1, 24 hours, n=43 | 1.379 (2.1969)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 1.503 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 57, 0.5 hours, n=31: number analyzed (Participants) | 31
  Day 57, 0.5 hours, n=31 | 7.760 (12.2768)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 10.507 (13.6474)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 20.254 (20.1125)
  Day 57, 3 hours, n=30: number analyzed (Participants) | 30
  Day 57, 3 hours, n=30 | 25.092 (20.7688)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 24.865 (18.7941)
  Day 57, 6 hours, n=31: number analyzed (Participants) | 31
  Day 57, 6 hours, n=31 | 21.749 (16.6572)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 11.419 (11.2821)
  Day 57, 12 hours, n=31: number analyzed (Participants) | 31
  Day 57, 12 hours, n=31 | 5.537 (9.1160)
  Day 57, 16 hours, n=30: number analyzed (Participants) | 30
  Day 57, 16 hours, n=30 | 3.613 (6.4974)
  Day 57, 24 hours, n=31: number analyzed (Participants) | 31
  Day 57, 24 hours, n=31 | 1.693 (2.9455)

16. Secondary Outcome: Plasma Concentrations of Metabolite GSK2506102
Description: Blood samples were collected at indicated time points for the concentrations of metabolite GSK25206102.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 1.862 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 1 hour, n=44: number analyzed (Participants) | 44
  Day 1, 1 hour, n=44 | 2.575 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 5.999 (5.9281)
  Day 1, 3 hours, n=44: number analyzed (Participants) | 44
  Day 1, 3 hours, n=44 | 7.047 (6.3772)
  Day 1, 4 hours, n=43: number analyzed (Participants) | 43
  Day 1, 4 hours, n=43 | 7.554 (6.0767)
  Day 1, 6 hours, n=43: number analyzed (Participants) | 43
  Day 1, 6 hours, n=43 | 8.564 (5.0888)
  Day 1, 8 hours, n=42: number analyzed (Participants) | 42
  Day 1, 8 hours, n=42 | 9.379 (3.9554)
  Day 1, 12 hours, n=40: number analyzed (Participants) | 40
  Day 1, 12 hours, n=40 | 8.658 (3.6930)
  Day 1, 16 hours, n=42: number analyzed (Participants) | 42
  Day 1, 16 hours, n=42 | 8.225 (3.7400)
  Day 1, 24 hours, n=42: number analyzed (Participants) | 42
  Day 1, 24 hours, n=42 | 7.024 (3.5347)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 1.126 (1.0181)
  Day 57, 0.5 hours, n=30: number analyzed (Participants) | 30
  Day 57, 0.5 hours, n=30 | 2.472 (2.2298)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 2.890 (2.4847)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 5.082 (4.1937)
  Day 57, 3 hours, n=31: number analyzed (Participants) | 31
  Day 57, 3 hours, n=31 | 7.688 (5.7677)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 9.474 (6.3929)
  Day 57, 6 hours, n=30: number analyzed (Participants) | 30
  Day 57, 6 hours, n=30 | 11.507 (5.3600)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 10.945 (4.9425)
  Day 57, 12 hours, n=31: number analyzed (Participants) | 31
  Day 57, 12 hours, n=31 | 10.286 (5.1703)
  Day 57, 16 hours, n=31: number analyzed (Participants) | 31
  Day 57, 16 hours, n=31 | 9.735 (5.1306)
  Day 57, 24 hours, n=32: number analyzed (Participants) | 32
  Day 57, 24 hours, n=32 | 8.449 (3.7371)

17. Secondary Outcome: Plasma Concentrations of Metabolite GSK2531398
Description: Blood samples were collected at indicated time points for the concentrations of metabolite GSK2531398.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 4.409 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 1 hour, n=44: number analyzed (Participants) | 44
  Day 1, 1 hour, n=44 | 6.139 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 13.779 (13.5109)
  Day 1, 3 hours, n=44: number analyzed (Participants) | 44
  Day 1, 3 hours, n=44 | 15.087 (13.4427)
  Day 1, 4 hours, n=43: number analyzed (Participants) | 43
  Day 1, 4 hours, n=43 | 14.881 (12.5678)
  Day 1, 6 hours, n=43: number analyzed (Participants) | 43
  Day 1, 6 hours, n=43 | 14.907 (9.6957)
  Day 1, 8 hours, n=42: number analyzed (Participants) | 42
  Day 1, 8 hours, n=42 | 13.930 (7.4098)
  Day 1, 12 hours, n=40: number analyzed (Participants) | 40
  Day 1, 12 hours, n=40 | 9.784 (6.6328)
  Day 1, 16 hours, n=42: number analyzed (Participants) | 42
  Day 1, 16 hours, n=42 | 7.751 (5.9158)
  Day 1, 24 hours, n=42: number analyzed (Participants) | 42
  Day 1, 24 hours, n=42 | 4.687 (4.1099)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 1.246 (1.9695)
  Day 57, 0.5 hours, n=30: number analyzed (Participants) | 30
  Day 57, 0.5 hours, n=30 | 4.482 (5.7104)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 5.406 (5.8321)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 10.580 (10.1185)
  Day 57, 3 hours, n=31: number analyzed (Participants) | 31
  Day 57, 3 hours, n=31 | 15.191 (12.9991)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 17.904 (13.4024)
  Day 57, 6 hours, n=30: number analyzed (Participants) | 30
  Day 57, 6 hours, n=30 | 19.827 (11.4600)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 15.038 (11.0475)
  Day 57, 12 hours, n=31: number analyzed (Participants) | 31
  Day 57, 12 hours, n=31 | 10.292 (8.2309)
  Day 57, 16 hours, n=31: number analyzed (Participants) | 31
  Day 57, 16 hours, n=31 | 8.348 (7.1590)
  Day 57, 24 hours, n=32: number analyzed (Participants) | 32
  Day 57, 24 hours, n=32 | 5.334 (4.8807)

18. Secondary Outcome: Plasma Concentrations of Metabolite GSK2531401
Description: Blood samples were collected at indicated time points for the concentrations of metabolite GSK2531401.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 45
Nanograms per milliliter
  Day 1, Predose, n=45 | 0.000 (0.000)
  Day 1, 0.5 hours, n=43: number analyzed (Participants) | 43
  Day 1, 0.5 hours, n=43 | 2.927 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 1 hour, n=44: number analyzed (Participants) | 44
  Day 1, 1 hour, n=44 | 4.134 (NA) — NA indicates SD could not be calculated due to the high proportion of NQ values (>30% of values were imputed) which affected the SD.
  Day 1, 2 hours, n=43: number analyzed (Participants) | 43
  Day 1, 2 hours, n=43 | 11.013 (11.9279)
  Day 1, 3 hours, n=44: number analyzed (Participants) | 44
  Day 1, 3 hours, n=44 | 13.752 (14.0238)
  Day 1, 4 hours, n=43: number analyzed (Participants) | 43
  Day 1, 4 hours, n=43 | 15.497 (14.6142)
  Day 1, 6 hours, n=43: number analyzed (Participants) | 43
  Day 1, 6 hours, n=43 | 18.302 (13.9244)
  Day 1, 8 hours, n=42: number analyzed (Participants) | 42
  Day 1, 8 hours, n=42 | 21.139 (13.2221)
  Day 1, 12 hours, n=40: number analyzed (Participants) | 40
  Day 1, 12 hours, n=40 | 20.174 (11.6828)
  Day 1, 16 hours, n=42: number analyzed (Participants) | 42
  Day 1, 16 hours, n=42 | 20.127 (12.1374)
  Day 1, 24 hours, n=42: number analyzed (Participants) | 42
  Day 1, 24 hours, n=42 | 18.143 (11.6065)
  Day 57, Predose, n=31: number analyzed (Participants) | 31
  Day 57, Predose, n=31 | 2.448 (2.0199)
  Day 57, 0.5 hours, n=31: number analyzed (Participants) | 31
  Day 57, 0.5 hours, n=31 | 4.486 (3.9244)
  Day 57, 1 hour, n=31: number analyzed (Participants) | 31
  Day 57, 1 hour, n=31 | 5.480 (5.0425)
  Day 57, 2 hours, n=30: number analyzed (Participants) | 30
  Day 57, 2 hours, n=30 | 9.015 (8.4201)
  Day 57, 3 hours, n=31: number analyzed (Participants) | 31
  Day 57, 3 hours, n=31 | 14.027 (12.7046)
  Day 57, 4 hours, n=32: number analyzed (Participants) | 32
  Day 57, 4 hours, n=32 | 17.722 (14.2802)
  Day 57, 6 hours, n=30: number analyzed (Participants) | 30
  Day 57, 6 hours, n=30 | 24.285 (15.7868)
  Day 57, 8 hours, n=31: number analyzed (Participants) | 31
  Day 57, 8 hours, n=31 | 25.557 (16.2248)
  Day 57, 12 hours, n=31: number analyzed (Participants) | 31
  Day 57, 12 hours, n=31 | 25.288 (15.7597)
  Day 57, 16 hours, n=31: number analyzed (Participants) | 31
  Day 57, 16 hours, n=31 | 24.881 (15.3688)
  Day 57, 24 hours, n=32: number analyzed (Participants) | 32
  Day 57, 24 hours, n=32 | 21.914 (12.9806)

19. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Daprodustat, GSK2391220, GSK2487818, GSK2506102, GSK2506104, GSK2531398 and GSK2531401
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of daprodustat and its metabolites GSK2391220, GSK2487818, GSK2506102, GSK2506104, GSK2531398 and GSK2531401. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 44
Nanograms per milliliter
  Daprodustat, Day 1, n=44 | 218.841 (187.869)
  Daprodustat, Day 57, n=32: number analyzed (Participants) | 32
  Daprodustat, Day 57, n=32 | 163.795 (330.249)
  GSK2391220, Day 1, n=44 | 39.506 (66.816)
  GSK2391220, Day 57, n=32: number analyzed (Participants) | 32
  GSK2391220, Day 57, n=32 | 44.703 (57.029)
  GSK2487818, Day 1, n=44 | 26.678 (79.992)
  GSK2487818, Day 57, n=32: number analyzed (Participants) | 32
  GSK2487818, Day 57, n=32 | 24.846 (117.570)
  GSK2506102, Day 1, n=44 | 9.933 (62.188)
  GSK2506102, Day 57, n=32: number analyzed (Participants) | 32
  GSK2506102, Day 57, n=32 | 12.114 (46.563)
  GSK2506104, Day 1, n=44 | 43.169 (61.558)
  GSK2506104, Day 57, n=32: number analyzed (Participants) | 32
  GSK2506104, Day 57, n=32 | 51.643 (48.087)
  GSK2531398, Day 1, n=44 | 18.454 (67.277)
  GSK2531398, Day 57, n=32: number analyzed (Participants) | 32
  GSK2531398, Day 57, n=32 | 20.362 (67.040)
  GSK2531401, Day 1, n=44 | 18.335 (96.906)
  GSK2531401, Day 57, n=32: number analyzed (Participants) | 32
  GSK2531401, Day 57, n=32 | 23.337 (75.801)

20. Secondary Outcome: Time of Occurrence of Cmax (Tmax) of Daprodustat, GSK2391220, GSK2487818, GSK2506102, GSK2506104, GSK2531398 and GSK2531401
Description: as for outcome 19
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Daprodustat
Number analyzed (Participants) | 44
Hours
  Daprodustat, Day 1, n=44 | 2.000 [0.38 to 8.00]
  Daprodustat, Day 57, n=32: number analyzed (Participants) | 32
  Daprodustat, Day 57, n=32 | 2.000 [0.50 to 12.00]
  GSK2391220, Day 1, n=44 | 4.160 [0.50 to 16.00]
  GSK2391220, Day 57, n=32: number analyzed (Participants) | 32
  GSK2391220, Day 57, n=32 | 4.000 [0.50 to 16.00]
  GSK2487818, Day 1, n=44 | 3.090 [0.50 to 12.00]
  GSK2487818, Day 57, n=32: number analyzed (Participants) | 32
  GSK2487818, Day 57, n=32 | 4.000 [0.50 to 12.00]
  GSK2506102, Day 1, n=44 | 6.000 [0.50 to 24.00]
  GSK2506102, Day 57, n=32: number analyzed (Participants) | 32
  GSK2506102, Day 57, n=32 | 6.000 [2.00 to 24.00]
  GSK2506104, Day 1, n=44 | 6.000 [0.50 to 16.30]
  GSK2506104, Day 57, n=32: number analyzed (Participants) | 32
  GSK2506104, Day 57, n=32 | 5.990 [0.50 to 24.00]
  GSK2531398, Day 1, n=44 | 4.160 [0.50 to 24.00]
  GSK2531398, Day 57, n=32: number analyzed (Participants) | 32
  GSK2531398, Day 57, n=32 | 4.000 [0.50 to 16.00]
  GSK2531401, Day 1, n=44 | 8.015 [1.00 to 24.50]
  GSK2531401, Day 57, n=32: number analyzed (Participants) | 32
  GSK2531401, Day 57, n=32 | 8.000 [3.00 to 24.00]

21. Secondary Outcome: Terminal Phase Half-life (t1/2) of Daprodustat, GSK2391220, GSK2487818, GSK2506102, GSK2506104, GSK2531398 and GSK2531401
Description: as for outcome 19
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Daprodustat
Number analyzed (Participants) | 44
Hours
  Daprodustat, Day 1, n=22: number analyzed (Participants) | 22
  Daprodustat, Day 1, n=22 | 3.031 (40.320)
  Daprodustat, Day 57, n=10: number analyzed (Participants) | 10
  Daprodustat, Day 57, n=10 | 3.635 (26.884)
  GSK2391220, Day 1, n=9: number analyzed (Participants) | 9
  GSK2391220, Day 1, n=9 | 6.820 (22.096)
  GSK2391220, Day 57, n=4: number analyzed (Participants) | 4
  GSK2391220, Day 57, n=4 | 7.447 (7.539)
  GSK2487818, Day 1, n=20: number analyzed (Participants) | 20
  GSK2487818, Day 1, n=20 | 3.388 (22.165)
  GSK2487818, Day 57, n=13: number analyzed (Participants) | 13
  GSK2487818, Day 57, n=13 | 3.524 (32.634)
  GSK2506102, Day 1, n=1: number analyzed (Participants) | 1
  GSK2506102, Day 1, n=1 | 8.530 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.
  GSK2506102, Day 57, n=32: number analyzed (Participants) | 32
  GSK2506102, Day 57, n=32 | NA (NA) — NA indicates data were not analyzed for t1/2 as there were not enough data points collected for a terminal slope required to calculate t1/2.
  GSK2506104, Day 1, n=1: number analyzed (Participants) | 1
  GSK2506104, Day 1, n=1 | 6.150 (NA) — NA indicates geometric coefficient of variation could not be calculated for single participant.
  GSK2506104, Day 57, n=32: number analyzed (Participants) | 32
  GSK2506104, Day 57, n=32 | NA (NA) — NA indicates data were not analyzed for t1/2 as there were not enough data points collected for a terminal slope required to calculate t1/2.
  GSK2531398, Day 1, n=11: number analyzed (Participants) | 11
  GSK2531398, Day 1, n=11 | 5.582 (22.955)
  GSK2531398, Day 57, n=9: number analyzed (Participants) | 9
  GSK2531398, Day 57, n=9 | 6.182 (14.307)
  GSK2531401, Day 1, n=44 | NA (NA) — NA indicates data were not analyzed for t1/2 as there were not enough data points collected for a terminal slope required to calculate t1/2.
  GSK2531401, Day 57, n=32: number analyzed (Participants) | 32
  GSK2531401, Day 57, n=32 | NA (NA) — NA indicates data were not analyzed for t1/2 as there were not enough data points collected for a terminal slope required to calculate t1/2.

22. Secondary Outcome: Area Under Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) of Daprodustat, GSK2391220, GSK2487818, GSK2506102, GSK2506104, GSK2531398 and GSK2531401
Description: as for outcome 19
Time Frame: Pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 16 and 24 hours on Days 1 and 57
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Daprodustat
Number analyzed (Participants) | 42
Hour*nanograms per milliliter
  Daprodustat, Day 1, n=42 | 767.95 (125.63)
  Daprodustat, Day 57, n=28: number analyzed (Participants) | 28
  Daprodustat, Day 57, n=28 | 616.12 (168.05)
  GSK2391220, Day 1, n=42 | 483.12 (60.42)
  GSK2391220, Day 57, n=31: number analyzed (Participants) | 31
  GSK2391220, Day 57, n=31 | 516.59 (61.78)
  GSK2487818, Day 1, n=41: number analyzed (Participants) | 41
  GSK2487818, Day 1, n=41 | 177.39 (66.83)
  GSK2487818, Day 57, n=28: number analyzed (Participants) | 28
  GSK2487818, Day 57, n=28 | 171.09 (93.41)
  GSK2506102, Day 1, n=42 | 166.89 (52.93)
  GSK2506102, Day 57, n=31: number analyzed (Participants) | 31
  GSK2506102, Day 57, n=31 | 199.85 (44.33)
  GSK2506104, Day 1, n=42 | 662.23 (54.48)
  GSK2506104, Day 57, n=31: number analyzed (Participants) | 31
  GSK2506104, Day 57, n=31 | 756.39 (50.29)
  GSK2531398, Day 1, n=42 | 204.02 (59.48)
  GSK2531398, Day 57, n=31: number analyzed (Participants) | 31
  GSK2531398, Day 57, n=31 | 212.04 (66.63)
  GSK2531401, Day 1, n=42 | 334.86 (93.49)
  GSK2531401, Day 57, n=31: number analyzed (Participants) | 31
  GSK2531401, Day 57, n=31 | 430.10 (73.53)

23. Other Pre Specified Outcome: Number of Participants With Any Serious Adverse Events (SAEs)
Description: Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly or birth defect or any other situation according to medical or scientific judgment was categorized as SAE.
Time Frame: Up to Week 10
Population: Safety Population comprises of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Participants | 10 | 5

24. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Common (>=2%) Non-serious Adverse Events (Non-SAEs)
Description: An AE is any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with study treatment. Number of participants with treatment emergent common (>=2% non-SAEs in each arm) non-SAEs has been presented.
Time Frame: Up to Week 8
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Participants | 10 | 4

25. Other Pre Specified Outcome: Number of Participants Who Discontinued the Study Treatment
Description: Number of participants who discontinued the study treatment due to any reason are presented. The reasons for discontinuation included adverse events, protocol specified withdrawal criteria met, physician decision and withdrawal by participant.
Time Frame: Up to Week 10
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Participants
  Adverse event | 2 | 2
  Protocol-specified withdrawal criteria met | 7 | 4
  Physician decision | 1 | 1
  Withdrawal by participant | 3 | 0

26. Other Pre Specified Outcome: Absolute Values for Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including albumin and protein. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: Safety Population. Only those participants with data available at specified time points has been presented (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Grams per liter
  Albumin, Baseline (Day1), n=45, 43 | 41.2 (3.42) | 40.5 (4.21)
  Albumin, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Albumin, Day 29, n=37, 40 | 39.1 (3.58) | 38.3 (4.02)
  Albumin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Albumin, Day 57, n=31, 35 | 41.4 (4.35) | 40.9 (4.83)
  Albumin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Albumin, Week 10, n=39, 38 | 38.7 (3.20) | 38.0 (5.19)
  Protein, Baseline (Day 1), n=45, 43 | 72.3 (7.27) | 72.6 (8.30)
  Protein, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Protein, Day 29, n=37, 40 | 69.4 (5.67) | 68.0 (7.92)
  Protein, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Protein, Day 57, n=31, 35 | 74.0 (7.51) | 73.1 (8.59)
  Protein, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Protein, Week 10, n=39, 38 | 67.5 (5.67) | 67.8 (7.79)

27. Other Pre Specified Outcome: Absolute Values for Clinical Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALP, ALT and AST. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
International units per liter
  ALP, Baseline (Day1), n=45, 43 | 100.9 (51.78) | 100.0 (40.47)
  ALP, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  ALP, Day 29, n=37, 40 | 104.4 (49.97) | 95.7 (37.28)
  ALP, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  ALP, Day 57, n=31, 35 | 109.0 (48.09) | 101.7 (37.81)
  ALP, Week 10, n=42, 41: number analyzed (Participants) | 42 | 41
  ALP, Week 10, n=42, 41 | 98.3 (54.64) | 98.8 (40.03)
  ALT, Baseline (Day 1), n=45, 43 | 13.8 (6.74) | 15.0 (6.97)
  ALT, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  ALT, Day 29, n=37, 40 | 10.4 (3.95) | 12.0 (5.80)
  ALT, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  ALT, Day 57, n=31, 35 | 11.0 (5.75) | 12.9 (5.07)
  ALT, Week 10, n=42, 41: number analyzed (Participants) | 42 | 41
  ALT, Week 10, n=42, 41 | 10.6 (4.71) | 12.3 (7.01)
  AST, Baseline (Day 1), n=45, 43 | 16.8 (6.63) | 17.0 (6.07)
  AST, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  AST, Day 29, n=37, 40 | 13.2 (4.76) | 13.7 (5.68)
  AST, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  AST, Day 57, n=31, 35 | 14.9 (5.12) | 15.2 (4.23)
  AST, Week 10, n=42, 41: number analyzed (Participants) | 42 | 41
  AST, Week 10, n=42, 41 | 14.0 (5.18) | 15.2 (10.86)

28. Other Pre Specified Outcome: Absolute Values for Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Indirect (Indrt) Bilirubin
Description: Blood samples were collected for the analysis of clinical chemistry parameters including direct bilirubin, total bilirubin and Indrt bilirubin. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Micromoles per liter
  Direct bilirubin,Baseline(Day1),n=45,43 | 2.0 (1.24) | 1.8 (1.17)
  Direct bilirubin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Direct bilirubin, Day 29, n=37, 39 | 1.9 (1.05) | 1.7 (1.23)
  Direct bilirubin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Direct bilirubin, Day 57, n=31, 35 | 1.9 (1.21) | 1.8 (1.35)
  Direct bilirubin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Direct bilirubin, Week 10, n=39, 38 | 1.8 (0.89) | 1.7 (1.09)
  Total bilirubin, Baseline (Day 1),n=45,43 | 8.6 (3.07) | 7.7 (3.25)
  Total bilirubin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Total bilirubin, Day 29, n=37, 39 | 7.1 (2.19) | 7.2 (1.93)
  Total bilirubin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Total bilirubin, Day 57, n=31, 35 | 9.0 (3.86) | 8.6 (2.69)
  Total bilirubin, Week 10, n=42, 41: number analyzed (Participants) | 42 | 41
  Total bilirubin, Week 10, n=42, 41 | 7.7 (2.29) | 7.0 (2.20)
  Indrt bilirubin, Baseline (Day 1), n=45,43 | 6.6 (2.28) | 6.0 (2.74)
  Indrt bilirubin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Indrt bilirubin, Day 29, n=37, 39 | 5.2 (1.79) | 5.4 (1.89)
  Indrt bilirubin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Indrt bilirubin, Day 57, n=31, 35 | 7.0 (3.30) | 6.9 (2.02)
  Indrt bilirubin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Indrt bilirubin, Week 10, n=39, 38 | 5.9 (2.08) | 5.3 (1.83)

29. Other Pre Specified Outcome: Absolute Values for Clinical Chemistry Parameters: Calcium Corrected for Albumin (CCA), Glucose, Potassium, Phosphate and Sodium
Description: Blood samples were collected for the analysis of clinical chemistry parameters including CCA, glucose, potassium, phosphate and sodium. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Millimoles per liter
  CCA, Baseline (Day 1),n=45,43 | 2.254 (0.1147) | 2.266 (0.1341)
  CCA, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  CCA, Day 29, n=37, 40 | 2.242 (0.1692) | 2.242 (0.1479)
  CCA, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  CCA, Day 57, n=31, 35 | 2.240 (0.1389) | 2.265 (0.1086)
  CCA, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  CCA, Week 10, n=39, 38 | 2.227 (0.1599) | 2.232 (0.1644)
  Glucose, Baseline (Day 1), n=45,43 | 7.40 (2.794) | 7.67 (3.504)
  Glucose, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Glucose, Day 29, n=37, 40 | 8.28 (4.234) | 7.35 (2.362)
  Glucose, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Glucose, Day 57, n=31, 35 | 7.27 (2.419) | 7.01 (2.690)
  Glucose, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Glucose, Week 10, n=39, 38 | 7.98 (3.020) | 7.36 (2.948)
  Potassium, Baseline (Day 1), n=45,43 | 3.99 (0.509) | 4.06 (0.788)
  Potassium, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Potassium, Day 29, n=37, 40 | 4.39 (0.769) | 4.60 (0.765)
  Potassium, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Potassium, Day 57, n=31, 35 | 3.81 (0.414) | 4.01 (0.663)
  Potassium, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Potassium, Week 10, n=39, 38 | 4.66 (0.639) | 4.65 (0.693)
  Phosphate, Baseline (Day 1), n=45,43 | 1.129 (0.4792) | 1.242 (0.5758)
  Phosphate, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Phosphate, Day 29, n=37, 40 | 1.455 (0.5207) | 1.761 (0.6297)
  Phosphate, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Phosphate, Day 57, n=31, 35 | 0.953 (0.2523) | 1.274 (0.6260)
  Phosphate, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Phosphate, Week 10, n=39, 38 | 1.629 (0.560) | 1.849 (0.5431)
  Sodium, Baseline (Day 1), n=45,43 | 137.9 (2.64) | 138.0 (2.58)
  Sodium, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Sodium, Day 29, n=37, 40 | 137.8 (2.41) | 138.4 (2.84)
  Sodium, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Sodium, Day 57, n=31, 35 | 137.7 (2.22) | 138.6 (2.74)
  Sodium, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Sodium, Week 10, n=39, 38 | 137.9 (2.28) | 138.6 (2.77)

30. Other Pre Specified Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including albumin and protein. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 40
Grams per liter
  Albumin, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Albumin, Day 29, n=37, 40 | -2.2 (3.67) | -2.4 (3.42)
  Albumin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Albumin, Day 57, n=31, 35 | 0.4 (3.60) | 0.5 (3.16)
  Albumin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Albumin, Week 10, n=39, 38 | -2.9 (3.10) | -2.4 (3.93)
  Protein, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Protein, Day 29, n=37, 40 | -3.7 (6.41) | -4.7 (6.03)
  Protein, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Protein, Day 57, n=31, 35 | 1.2 (6.44) | 0.7 (5.64)
  Protein, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Protein, Week 10, n=39, 38 | -5.2 (5.90) | -4.9 (5.69)

31. Other Pre Specified Outcome: Change From Baseline Values for Clinical Chemistry Parameters: ALP, ALT and AST
Description: Blood samples were collected for the analysis of clinical chemistry parameters including ALP, ALT and AST. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 42 | 41
International units per liter
  ALP, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  ALP, Day 29, n=37, 40 | -3.4 (19.56) | -5.3 (27.57)
  ALP, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  ALP, Day 57, n=31, 35 | 0.5 (23.21) | 3.4 (17.93)
  ALP, Week 10, n=42, 41 | -4.5 (29.46) | -1.9 (25.70)
  ALT, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  ALT, Day 29, n=37, 40 | -3.2 (5.74) | -2.6 (6.36)
  ALT, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  ALT, Day 57, n=31, 35 | -3.1 (7.93) | -1.9 (5.93)
  ALT, Week 10, n=42, 41 | -3.3 (7.31) | -2.8 (4.96)
  AST, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  AST, Day 29, n=37, 40 | -3.2 (4.90) | -3.0 (5.38)
  AST, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  AST, Day 57, n=31, 35 | -2.1 (6.10) | -1.9 (4.60)
  AST, Week 10, n=42, 41 | -3.3 (6.10) | -2.0 (9.11)

32. Other Pre Specified Outcome: Change From Baseline Values for Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin and Indrt. Bilirubin
Description: Blood samples were collected for the analysis of clinical chemistry parameters including direct bilirubin, total bilirubin and indrt. bilirubin. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 42 | 41
Micromoles per liter
  Direct bilirubin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Direct bilirubin, Day 29, n=37, 39 | -0.1 (1.05) | -0.1 (1.69)
  Direct bilirubin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Direct bilirubin, Day 57, n=31, 35 | -0.1 (1.21) | -0.1 (1.37)
  Direct bilirubin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Direct bilirubin, Week 10, n=39, 38 | -0.3 (1.14) | -0.1 (1.18)
  Total bilirubin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Total bilirubin, Day 29, n=37, 39 | -1.5 (2.19) | -0.8 (3.10)
  Total bilirubin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Total bilirubin, Day 57, n=31, 35 | 0.6 (2.74) | 0.7 (2.70)
  Total bilirubin, Week 10, n=42, 41 | -1.0 (2.62) | -0.8 (2.23)
  Indrt bilirubin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Indrt bilirubin, Day 29, n=37, 39 | -1.4 (2.06) | -0.7 (2.92)
  Indrt bilirubin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Indrt bilirubin, Day 57, n=31, 35 | 0.6 (2.80) | 0.9 (2.80)
  Indrt bilirubin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Indrt bilirubin, Week 10, n=39, 38 | -0.8 (2.28) | -0.5 (2.01)

33. Other Pre Specified Outcome: Change From Baseline Values for Clinical Chemistry Parameters: CCA, Glucose, Potassium, Phosphate and Sodium
Description: Blood samples were collected for the analysis of clinical chemistry parameters including CCA, glucose, potassium, phosphate and sodium. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 40
Millimoles per liter
  CCA, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  CCA, Day 29, n=37, 40 | 0.000 (0.1384) | -0.021 (0.1699)
  CCA, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  CCA, Day 57, n=31, 35 | 0.004 (0.1344) | -0.000 (0.1450)
  CCA, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  CCA, Week 10, n=39, 38 | -0.010 (0.1693) | -0.033 (0.1284)
  Glucose, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Glucose, Day 29, n=37, 40 | 0.75 (4.331) | -0.48 (3.771)
  Glucose, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Glucose, Day 57, n=31, 35 | -0.45 (2.403) | -0.83 (2.684)
  Glucose, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Glucose, Week 10, n=39, 38 | 0.62 (3.001) | -0.18 (2.916)
  Potassium, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Potassium, Day 29, n=37, 40 | 0.45 (0.790) | 0.53 (0.863)
  Potassium, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Potassium, Day 57, n=31, 35 | -0.14 (0.512) | -0.04 (0.696)
  Potassium, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Potassium, Week 10, n=39, 38 | 0.67 (0.694) | 0.58 (0.746)
  Phosphate, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Phosphate, Day 29, n=37, 40 | 0.389 (0.6876) | 0.513 (0.7270)
  Phosphate, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Phosphate, Day 57, n=31, 35 | -0.123 (0.4624) | 0.004 (0.5274)
  Phosphate, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Phosphate, Week 10, n=39, 38 | 0.505 (0.7016) | 0.599 (0.6723)
  Sodium, Day 29, n=37, 40: number analyzed (Participants) | 37 | 40
  Sodium, Day 29, n=37, 40 | -0.1 (3.25) | 0.3 (3.22)
  Sodium, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Sodium, Day 57, n=31, 35 | 0.2 (2.47) | 0.6 (2.71)
  Sodium, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Sodium, Week 10, n=39, 38 | -0.2 (2.41) | 0.5 (2.53)

34. Other Pre Specified Outcome: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 42
10^9 cells per liter
  Basophils, Baseline (Day 1), n=45, 41: number analyzed (Participants) | 45 | 41
  Basophils, Baseline (Day 1), n=45, 41 | 0.050 (0.0295) | 0.044 (0.0255)
  Basophils, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Basophils, Day 29, n=37, 39 | 0.045 (0.0301) | 0.054 (0.0312)
  Basophils, Day 57, n=30, 35: number analyzed (Participants) | 30 | 35
  Basophils, Day 57, n=30, 35 | 0.049 (0.0349) | 0.045 (0.0243)
  Basophils, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Basophils, Week 10, n=39, 38 | 0.044 (0.0261) | 0.054 (0.0284)
  Eosinophils, Baseline (Day 1), n=45, 41: number analyzed (Participants) | 45 | 41
  Eosinophils, Baseline (Day 1), n=45, 41 | 0.196 (0.1520) | 0.229 (0.2324)
  Eosinophils, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Eosinophils, Day 29, n=37, 39 | 0.238 (0.2301) | 0.191 (0.1551)
  Eosinophils, Day 57, n=30, 35: number analyzed (Participants) | 30 | 35
  Eosinophils, Day 57, n=30, 35 | 0.218 (0.1811) | 0.160 (0.1505)
  Eosinophils, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Eosinophils, Week 10, n=39, 38 | 0.231 (0.1918) | 0.184 (0.1167)
  Lymphocytes, Baseline (Day 1), n=45, 41: number analyzed (Participants) | 45 | 41
  Lymphocytes, Baseline (Day 1), n=45, 41 | 1.257 (0.3926) | 1.307 (0.6305)
  Lymphocytes, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Lymphocytes, Day 29, n=37, 39 | 1.385 (0.5446) | 1.436 (0.5798)
  Lymphocytes, Day 57, n=30, 35: number analyzed (Participants) | 30 | 35
  Lymphocytes, Day 57, n=30, 35 | 1.209 (0.5062) | 1.225 (0.6698)
  Lymphocytes, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Lymphocytes, Week 10, n=39, 38 | 1.367 (0.5559) | 1.408 (0.6788)
  Monocytes, Baseline (Day 1), n=45, 41: number analyzed (Participants) | 45 | 41
  Monocytes, Baseline (Day 1), n=45, 41 | 0.398 (0.1471) | 0.408 (0.1752)
  Monocytes, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Monocytes, Day 29, n=37, 39 | 0.442 (0.1664) | 0.460 (0.1812)
  Monocytes, Day 57, n=30, 35: number analyzed (Participants) | 30 | 35
  Monocytes, Day 57, n=30, 35 | 0.432 (0.1621) | 0.448 (0.2204)
  Monocytes, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Monocytes, Week 10, n=39, 38 | 0.469 (0.1640) | 0.443 (0.1773)
  Neutrophils, Baseline (Day 1), n=45, 41: number analyzed (Participants) | 45 | 41
  Neutrophils, Baseline (Day 1), n=45, 41 | 4.091 (1.6571) | 4.053 (1.4574)
  Neutrophils, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Neutrophils, Day 29, n=37, 39 | 4.319 (1.3509) | 4.242 (1.5623)
  Neutrophils, Day 57, n=30, 35: number analyzed (Participants) | 30 | 35
  Neutrophils, Day 57, n=30, 35 | 4.381 (1.9926) | 4.377 (1.6450)
  Neutrophils, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Neutrophils, Week 10, n=39, 38 | 4.250 (1.8123) | 4.369 (1.7463)
  Platelets, Baseline (Day 1), n=45, 42 | 188.5 (67.64) | 193.8 (70.03)
  Platelets, Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Platelets, Day 29, n=37, 38 | 195.2 (66.55) | 222.1 (82.78)
  Platelets, Day 57, n=30, 34: number analyzed (Participants) | 30 | 34
  Platelets, Day 57, n=30, 34 | 207.8 (95.04) | 213.5 (67.33)
  Platelets, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Platelets, Week 10, n=39, 38 | 209.3 (75.61) | 229.5 (78.29)
  Leukocytes, Baseline (Day 1), n=45, 41: number analyzed (Participants) | 45 | 41
  Leukocytes, Baseline (Day 1), n=45, 41 | 6.00 (1.923) | 6.04 (1.897)
  Leukocytes, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Leukocytes, Day 29, n=37, 39 | 6.43 (1.678) | 6.38 (2.145)
  Leukocytes, Day 57, n=30, 35: number analyzed (Participants) | 30 | 35
  Leukocytes, Day 57, n=30, 35 | 6.29 (2.363) | 6.25 (2.044)
  Leukocytes, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Leukocytes, Week 10, n=39, 38 | 6.35 (2.178) | 6.45 (2.297)

35. Other Pre Specified Outcome: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 42
Proportion of red blood cells in blood
  Baseline (Day 1), n=45, 42 | 0.3133 (0.03111) | 0.3242 (0.03046)
  Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Day 29, n=37, 39 | 0.3066 (0.03195) | 0.3113 (0.03307)
  Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Day 57, n=31, 35 | 0.3196 (0.03046) | 0.3397 (0.02476)
  Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Week 10, n=39, 38 | 0.3050 (0.03743) | 0.3209 (0.03375)

36. Other Pre Specified Outcome: Absolute Values for Hematology Parameters: Erythrocytes and Reticulocytes
Description: Blood samples were collected for the analysis of hematology parameters: erythrocytes and reticulocytes. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 42
10^12 cells per liter
  Erythrocytes, Baseline (Day 1), n=45, 42 | 3.31 (0.378) | 3.45 (0.388)
  Erythrocytes, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Erythrocytes, Day 29, n=37, 39 | 3.20 (0.361) | 3.27 (0.499)
  Erythrocytes, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Erythrocytes, Day 57, n=31, 35 | 3.34 (0.393) | 3.53 (0.357)
  Erythrocytes, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Erythrocytes, Week 10, n=39, 38 | 3.13 (0.388) | 3.38 (0.470)
  Reticulocytes, Baseline (Day 1), n=45, 42 | 0.0302 (0.01536) | 0.0401 (0.02614)
  Reticulocytes, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Reticulocytes, Day 29, n=37, 39 | 0.0486 (0.01676) | 0.0733 (0.03493)
  Reticulocytes, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Reticulocytes, Day 57, n=31, 35 | 0.0489 (0.01681) | 0.0627 (0.03344)
  Reticulocytes, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Reticulocytes, Week 10, n=39, 38 | 0.0613 (0.03932) | 0.0566 (0.03060)

37. Other Pre Specified Outcome: Absolute Values for Hematology Parameters: Hemoglobin and Erythrocyte Mean Corpusclar Hemoglobin Concentration ( Ery. MCHC)
Description: Blood samples were collected for the analysis of hematology parameters: hemoglobin and ery.MCHC. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 42
Grams per liter
  Hemoglobin, Baseline (Day 1), n=45, 42 | 102.2 (9.15) | 104.5 (8.83)
  Hemoglobin, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Hemoglobin, Day 29, n=37, 39 | 100.2 (10.01) | 99.7 (9.63)
  Hemoglobin, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Hemoglobin, Day 57, n=31, 35 | 105.2 (9.61) | 107.9 (6.01)
  Hemoglobin, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Hemoglobin, Week 10, n=39, 38 | 99.6 (12.44) | 102.9 (10.54)
  ery.MCHC, Baseline (Day 1), n=45, 42 | 326.7 (9.01) | 322.6 (8.41)
  ery.MCHC, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  ery.MCHC, Day 29, n=37, 39 | 327.1 (6.57) | 320.8 (11.50)
  ery.MCHC, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  ery.MCHC, Day 57, n=31, 35 | 329.0 (6.62) | 318.3 (15.46)
  ery.MCHC, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  ery.MCHC, Week 10, n=39, 38 | 326.7 (9.26) | 320.6 (9.17)

38. Other Pre Specified Outcome: Absolute Values for Hematology Parameter: Ery. Mean Corpuscular Hemoglobin (MCH) and Reticulocyte Corpuscular Hemoglobin Content (CHr)
Description: Blood samples were collected for the analysis of hematology parameter: ery.MCH and CHr. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Picograms
  ery. MCH, Baseline (Day 1), n=45, 42: number analyzed (Participants) | 45 | 42
  ery. MCH, Baseline (Day 1), n=45, 42 | 31.03 (2.295) | 30.57 (2.880)
  ery. MCH, Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  ery. MCH, Day 29, n=37, 39 | 31.56 (2.302) | 30.83 (3.051)
  ery. MCH, Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  ery. MCH, Day 57, n=31, 35 | 31.75 (2.312) | 30.88 (3.140)
  ery. MCH, Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  ery. MCH, Week 10, n=39, 38 | 31.96 (2.246) | 30.66 (2.823)
  CHr, Baseline (Day 1), n=45, 43 | 30.70 (1.730) | 29.97 (2.088)
  CHr, Day 29, n=36, 40: number analyzed (Participants) | 36 | 40
  CHr, Day 29, n=36, 40 | 30.55 (1.799) | 30.19 (2.242)
  CHr, Day 57, n=32, 36: number analyzed (Participants) | 32 | 36
  CHr, Day 57, n=32, 36 | 30.71 (1.852) | 29.85 (2.462)
  CHr, Week 10, n=39, 39: number analyzed (Participants) | 39 | 39
  CHr, Week 10, n=39, 39 | 30.55 (2.116) | 29.76 (2.079)

39. Other Pre Specified Outcome: Absolute Values for Hematology Parameter: Ery. Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of hematology parameter: ery.MCV. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 42
Femtoliters
  Baseline (Day 1), n=45, 42 | 95.0 (6.33) | 94.8 (8.37)
  Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Day 29, n=37, 39 | 96.5 (6.92) | 96.2 (8.76)
  Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Day 57, n=31, 35 | 96.5 (7.18) | 97.1 (9.04)
  Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Week 10, n=39, 38 | 97.9 (6.61) | 95.7 (8.37)

40. Other Pre Specified Outcome: Absolute Values for Hematology Parameter: Erythrocyte Distribution Width
Description: Blood samples were collected for the analysis of hematology parameter: erythrocyte distribution width. Baseline value (Day1) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 42
Percentage of width
  Baseline (Day 1), n=45, 42 | 16.06 (1.618) | 15.71 (1.917)
  Day 29, n=37, 39: number analyzed (Participants) | 37 | 39
  Day 29, n=37, 39 | 16.52 (1.802) | 16.75 (2.230)
  Day 57, n=31, 35: number analyzed (Participants) | 31 | 35
  Day 57, n=31, 35 | 16.11 (1.476) | 16.67 (2.034)
  Week 10, n=39, 38: number analyzed (Participants) | 39 | 38
  Week 10, n=39, 38 | 16.42 (2.036) | 16.45 (1.696)

41. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected for the analysis of hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 37
10^9 cells per liter
  Basophils, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Basophils, Day 29, n=37, 37 | -0.007 (0.0317) | 0.010 (0.0329)
  Basophils, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Basophils, Day 57, n=30, 33 | -0.002 (0.0331) | 0.004 (0.0335)
  Basophils, Week 10, n=39, 36: number analyzed (Participants) | 39 | 36
  Basophils, Week 10, n=39, 36 | -0.004 (0.0349) | 0.009 (0.0323)
  Eosinophils, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Eosinophils, Day 29, n=37, 37 | 0.040 (0.1717) | -0.039 (0.1728)
  Eosinophils, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Eosinophils, Day 57, n=30, 33 | 0.016 (0.1513) | -0.038 (0.1202)
  Eosinophils, Week 10, n=39, 36: number analyzed (Participants) | 39 | 36
  Eosinophils, Week 10, n=39, 36 | 0.042 (0.1435) | -0.036 (0.1702)
  Lymphocytes, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Lymphocytes, Day 29, n=37, 37 | 0.095 (0.3613) | 0.102 (0.4154)
  Lymphocytes, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Lymphocytes, Day 57, n=30, 33 | -0.090 (0.3036) | -0.099 (0.3277)
  Lymphocytes, Week 10, n=39, 36: number analyzed (Participants) | 39 | 36
  Lymphocytes, Week 10, n=39, 36 | 0.103 (0.3893) | 0.078 (0.4660)
  Monocytes, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Monocytes, Day 29, n=37, 37 | 0.033 (0.1600) | 0.035 (0.1266)
  Monocytes, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Monocytes, Day 57, n=30, 33 | 0.024 (0.1621) | 0.025 (0.1543)
  Monocytes, Week 10, n=39, 36: number analyzed (Participants) | 39 | 36
  Monocytes, Week 10, n=39, 36 | 0.070 (0.1398) | 0.053 (0.1248)
  Neutrophils, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Neutrophils, Day 29, n=37, 37 | 0.071 (1.1706) | 0.061 (1.3382)
  Neutrophils, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Neutrophils, Day 57, n=30, 33 | 0.081 (1.2291) | 0.325 (1.1549)
  Neutrophils, Week 10, n=39, 36: number analyzed (Participants) | 39 | 36
  Neutrophils, Week 10, n=39, 36 | 0.218 (1.3096) | 0.181 (0.9586)
  Platelets, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Platelets, Day 29, n=37, 37 | 0.6 (31.12) | 22.7 (52.46)
  Platelets, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Platelets, Day 57, n=30, 33 | 13.9 (47.04) | 16.4 (39.51)
  Platelets, Week 10, n=39, 37 | 20.6 (36.08) | 26.3 (41.87)
  Leukocytes, Day 29, n=37, 37: number analyzed (Participants) | 37 | 37
  Leukocytes, Day 29, n=37, 37 | 0.23 (1.296) | 0.17 (1.555)
  Leukocytes, Day 57, n=30, 33: number analyzed (Participants) | 30 | 33
  Leukocytes, Day 57, n=30, 33 | 0.02 (1.456) | 0.21 (1.231)
  Leukocytes, Week 10, n=39, 36: number analyzed (Participants) | 39 | 36
  Leukocytes, Week 10, n=39, 36 | 0.42 (1.442) | 0.28 (1.220)

42. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 38
Proportion of red blood cells in blood
  Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Day 29, n=37, 38 | -0.0131 (0.03062) | -0.0136 (0.02614)
  Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  Day 57, n=31, 34 | -0.0016 (0.03717) | 0.0131 (0.03609)
  Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  Week 10, n=39, 37 | -0.0096 (0.04571) | -0.0054 (0.04944)

43. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameters: Erythrocytes and Reticulocytes
Description: Blood samples were collected for the analysis of hematology parameters: erythrocytes and reticulocytes. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 38
10^12 cells per liter
  Erythrocytes, Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Erythrocytes, Day 29, n=37, 38 | -0.17 (0.331) | -0.20 (0.273)
  Erythrocytes, Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  Erythrocytes, Day 57, n=31, 34 | -0.06 (0.410) | 0.04 (0.307)
  Erythrocytes, Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  Erythrocytes, Week 10, n=39, 37 | -0.18 (0.488) | -0.11 (0.497)
  Reticulocytes, Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Reticulocytes, Day 29, n=37, 38 | 0.0156 (0.01432) | 0.0315 (0.03821)
  Reticulocytes, Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  Reticulocytes, Day 57, n=31, 34 | 0.0169 (0.01709) | 0.0204 (0.02182)
  Reticulocytes, Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  Reticulocytes, Week 10, n=39, 37 | 0.0314 (0.04385) | 0.0159 (0.02321)

44. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameters: Hemoglobin and Ery. MCHC
Description: Blood samples were collected for the analysis of hematology parameters: hemoglobin and ery.MCHC. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 38
Grams per liter
  Hemoglobin, Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Hemoglobin, Day 29, n=37, 38 | -4.1 (9.35) | -5.1 (8.21)
  Hemoglobin, Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  Hemoglobin, Day 57, n=31, 34 | 0.5 (10.60) | 2.5 (8.54)
  Hemoglobin, Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  Hemoglobin, Week 10, n=39, 37 | -3.2 (14.35) | -1.8 (14.46)
  ery.MCHC, Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  ery.MCHC, Day 29, n=37, 38 | 0.3 (8.41) | -2.0 (10.38)
  ery.MCHC, Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  ery.MCHC, Day 57, n=31, 34 | 2.3 (8.83) | -4.4 (14.46)
  ery.MCHC, Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  ery.MCHC, Week 10, n=39, 37 | -0.6 (9.37) | -0.8 (11.20)

45. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameters: Ery. MCH and CHr
Description: Blood samples were collected for the analysis of hematology parameter: ery.MCH and CHr. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 40
Picograms
  ery. MCH, Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  ery. MCH, Day 29, n=37, 38 | 0.39 (0.676) | 0.40 (0.672)
  ery. MCH, Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  ery. MCH, Day 57, n=31, 34 | 0.70 (1.161) | 0.49 (0.871)
  ery. MCH, Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  ery. MCH, Week 10, n=39, 37 | 0.78 (1.249) | 0.38 (1.000)
  CHr, Day 29, n=36, 40: number analyzed (Participants) | 36 | 40
  CHr, Day 29, n=36, 40 | -0.23 (0.937) | 0.20 (1.060)
  CHr, Day 57, n=32, 36: number analyzed (Participants) | 32 | 36
  CHr, Day 57, n=32, 36 | -0.12 (1.067) | -0.09 (1.617)
  CHr, Week 10, n=39, 39: number analyzed (Participants) | 39 | 39
  CHr, Week 10, n=39, 39 | -0.29 (1.696) | -0.03 (1.478)

46. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameter: Ery. MCV
Description: Blood samples were collected for the analysis of hematology parameter: ery.MCV. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 38
Femtoliters
  Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Day 29, n=37, 38 | 1.2 (2.47) | 1.8 (3.32)
  Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  Day 57, n=31, 34 | 1.5 (3.50) | 2.9 (3.54)
  Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  Week 10, n=39, 37 | 2.7 (4.80) | 1.4 (3.62)

47. Other Pre Specified Outcome: Change From Baseline Values for Hematology Parameter: Erythrocyte Distribution Width
Description: Blood samples were collected for the analysis of hematology parameter: erythrocyte distribution width. Baseline value (Day1) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1) and at Days 29, 57 and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 39 | 38
Percentage of width
  Day 29, n=37, 38: number analyzed (Participants) | 37 | 38
  Day 29, n=37, 38 | 0.38 (1.197) | 1.09 (1.435)
  Day 57, n=31, 34: number analyzed (Participants) | 31 | 34
  Day 57, n=31, 34 | 0.12 (1.262) | 0.85 (1.609)
  Week 10, n=39, 37: number analyzed (Participants) | 39 | 37
  Week 10, n=39, 37 | 0.35 (1.998) | 0.59 (1.650)

48. Other Pre Specified Outcome: Absolute Values for Electrocardiogram (ECG) Mean Heart Rate
Description: Full 12-lead ECGs were obtained in supine position using an ECG machine to measure mean heart rate. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1-predose) and at Day 1: 24 hours; Day 57: pre-dose; Day 57: 24 hours and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Beats per minute
  Baseline (Day 1-predose), n=45, 43 | 72.2 (9.52) | 73.6 (9.03)
  Day 1: 24 hours, n=40, 38: number analyzed (Participants) | 40 | 38
  Day 1: 24 hours, n=40, 38 | 71.6 (9.38) | 74.8 (9.42)
  Day 57: predose, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: predose, n=32, 36 | 71.2 (8.58) | 72.7 (9.47)
  Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 24 hours, n=32, 36 | 71.2 (8.22) | 75.1 (9.12)
  Week 10, n=39, 40: number analyzed (Participants) | 39 | 40
  Week 10, n=39, 40 | 72.3 (10.03) | 74.3 (9.53)

49. Other Pre Specified Outcome: Absolute Values for ECG Parameters: PR Interval, QRS Duration, QT Interval Corrected for Heart Rate (QTc) and QT Interval Corrected for Heart Rate Using Bazett's Formula (QTcB)
Description: Full 12-lead ECGs were obtained in supine position using an ECG machine to measure ECG parameters: PR interval, QRS duration, QTc interval and QTcB. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1-predose) and at Day 1: 24 hours; Day 57: pre-dose; Day 57: 24 hours and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Milliseconds
  PR interval, Baseline (Day 1-predose), n=45, 43 | 156.5 (30.81) | 160.5 (30.79)
  PR interval, Day 1: 24 hours, n=39, 38: number analyzed (Participants) | 39 | 38
  PR interval, Day 1: 24 hours, n=39, 38 | 158.1 (30.26) | 163.3 (34.38)
  PR interval, Day 57: predose, n=32, 35: number analyzed (Participants) | 32 | 35
  PR interval, Day 57: predose, n=32, 35 | 155.8 (27.69) | 152.1 (26.90)
  PR interval, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  PR interval, Day 57: 24 hours, n=32, 36 | 156.4 (29.83) | 160.3 (32.98)
  PR interval, Week 10, n=39, 40: number analyzed (Participants) | 39 | 40
  PR interval, Week 10, n=39, 40 | 162.5 (29.19) | 159.9 (31.16)
  QRS duration, Baseline (Day 1-predose), n=45, 43 | 106.2 (18.40) | 107.4 (16.22)
  QRS duration, Day 1: 24 hours, n=40, 38: number analyzed (Participants) | 40 | 38
  QRS duration, Day 1: 24 hours, n=40, 38 | 106.0 (17.31) | 107.4 (17.85)
  QRS duration, Day 57: predose, n=32, 36: number analyzed (Participants) | 32 | 36
  QRS duration, Day 57: predose, n=32, 36 | 106.7 (14.46) | 112.4 (21.89)
  QRS duration, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  QRS duration, Day 57: 24 hours, n=32, 36 | 106.4 (15.05) | 111.0 (20.75)
  QRS duration, Week 10, n=39, 40: number analyzed (Participants) | 39 | 40
  QRS duration, Week 10, n=39, 40 | 108.5 (15.56) | 109.1 (20.69)
  QTc interval, Baseline (Day 1-predose), n=9, 17: number analyzed (Participants) | 9 | 17
  QTc interval, Baseline (Day 1-predose), n=9, 17 | 440.6 (22.41) | 429.4 (27.49)
  QTc interval, Day 1: 24 hours, n=7, 11: number analyzed (Participants) | 7 | 11
  QTc interval, Day 1: 24 hours, n=7, 11 | 446.1 (18.94) | 424.7 (27.73)
  QTc interval, Day 57: predose, n=5, 8: number analyzed (Participants) | 5 | 8
  QTc interval, Day 57: predose, n=5, 8 | 452.8 (13.92) | 436.1 (21.72)
  QTc interval, Day 57: 24 hours, n=5, 8: number analyzed (Participants) | 5 | 8
  QTc interval, Day 57: 24 hours, n=5, 8 | 430.6 (14.84) | 431.8 (31.98)
  QTc interval, Week 10, n=6, 10: number analyzed (Participants) | 6 | 10
  QTc interval, Week 10, n=6, 10 | 438.8 (13.01) | 428.3 (31.87)
  QTcB, Baseline (Day 1-predose), n=45, 43 | 448.0 (40.17) | 445.6 (31.00)
  QTcB, Day 1: 24 hours, n=40, 38: number analyzed (Participants) | 40 | 38
  QTcB, Day 1: 24 hours, n=40, 38 | 438.9 (35.02) | 439.3 (25.64)
  QTcB, Day 57: predose, n=32, 36: number analyzed (Participants) | 32 | 36
  QTcB, Day 57: predose, n=32, 36 | 442.3 (38.12) | 449.1 (32.58)
  QTcB, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  QTcB, Day 57: 24 hours, n=32, 36 | 437.4 (33.58) | 442.0 (37.61)
  QTcB, Week 10, n=39, 39: number analyzed (Participants) | 39 | 39
  QTcB, Week 10, n=39, 39 | 442.0 (37.28) | 441.6 (28.11)

50. Other Pre Specified Outcome: Change From Baseline Values for ECG Mean Heart Rate
Description: Full 12-lead ECGs were obtained in supine position using an ECG machine to measure mean heart rate. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1-predose) and at Day 1: 24 hours; Day 57: pre-dose; Day 57: 24 hours and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 40 | 40
Beats per minute
  Day 1: 24 hours, n=40, 38: number analyzed (Participants) | 40 | 38
  Day 1: 24 hours, n=40, 38 | -0.6 (6.85) | 0.8 (5.61)
  Day 57: predose, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: predose, n=32, 36 | -1.6 (7.25) | 0.1 (8.22)
  Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 24 hours, n=32, 36 | -1.7 (6.58) | 2.5 (8.21)
  Week 10, n=39, 40: number analyzed (Participants) | 39 | 40
  Week 10, n=39, 40 | -0.1 (9.01) | 0.4 (8.86)

51. Other Pre Specified Outcome: Change From Baseline Values for ECG Parameters: PR Interval, QRS Duration, QTc and QTcB
Description: Full 12-lead ECGs were obtained in supine position using an ECG machine to measure ECG parameters: PR interval, QRS duration, QTc interval and QTcB. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1-predose) and at Day 1: 24 hours; Day 57: pre-dose; Day 57: 24 hours and Week 10
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 40 | 40
Milliseconds
  PR interval, Day 1: 24 hours, n=39, 38: number analyzed (Participants) | 39 | 38
  PR interval, Day 1: 24 hours, n=39, 38 | 3.0 (11.02) | 1.9 (11.16)
  PR interval, Day 57: predose, n=32, 35: number analyzed (Participants) | 32 | 35
  PR interval, Day 57: predose, n=32, 35 | 0.2 (17.58) | -3.9 (11.34)
  PR interval, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  PR interval, Day 57: 24 hours, n=32, 36 | 0.8 (15.89) | 1.8 (13.03)
  PR interval, Week 10, n=39, 40: number analyzed (Participants) | 39 | 40
  PR interval, Week 10, n=39, 40 | 4.9 (15.21) | 1.2 (17.11)
  QRS duration, Day 1: 24 hours, n=40, 38: number analyzed (Participants) | 40 | 38
  QRS duration, Day 1: 24 hours, n=40, 38 | -0.5 (7.60) | 0.0 (4.73)
  QRS duration, Day 57: predose, n=32, 36: number analyzed (Participants) | 32 | 36
  QRS duration, Day 57: predose, n=32, 36 | 0.3 (9.53) | 2.8 (15.01)
  QRS duration, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  QRS duration, Day 57: 24 hours, n=32, 36 | 0.0 (11.13) | 1.4 (13.22)
  QRS duration, Week 10, n=39, 40: number analyzed (Participants) | 39 | 40
  QRS duration, Week 10, n=39, 40 | 0.8 (12.62) | 0.7 (18.38)
  QTc interval, Day 1: 24 hours, n=7, 11: number analyzed (Participants) | 7 | 11
  QTc interval, Day 1: 24 hours, n=7, 11 | 2.1 (14.59) | -9.4 (14.87)
  QTc interval, Day 57: predose, n=4, 8: number analyzed (Participants) | 4 | 8
  QTc interval, Day 57: predose, n=4, 8 | -6.3 (20.14) | 1.0 (5.71)
  QTc interval, Day 57: 24 hours, n=4, 8: number analyzed (Participants) | 4 | 8
  QTc interval, Day 57: 24 hours, n=4, 8 | -29.0 (31.89) | -3.4 (14.79)
  QTc interval, Week 10, n=6, 9: number analyzed (Participants) | 6 | 9
  QTc interval, Week 10, n=6, 9 | -6.7 (25.15) | -10.3 (11.74)
  QTcB, Day 1: 24 hours, n=40, 38: number analyzed (Participants) | 40 | 38
  QTcB, Day 1: 24 hours, n=40, 38 | -7.0 (24.13) | -3.1 (12.31)
  QTcB, Day 57: predose, n=32, 36: number analyzed (Participants) | 32 | 36
  QTcB, Day 57: predose, n=32, 36 | -7.0 (30.14) | 4.9 (12.36)
  QTcB, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  QTcB, Day 57: 24 hours, n=32, 36 | -12.0 (29.93) | -2.2 (23.15)
  QTcB, Week 10, n=39, 39: number analyzed (Participants) | 39 | 39
  QTcB, Week 10, n=39, 39 | -7.2 (35.84) | -3.0 (15.34)

52. Other Pre Specified Outcome: Absolute Values for Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs including SBP and DBP were measured in participants in a semi-supine position after 5 minutes rest. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1, predose) and at Day 1: 3, 12, 24 hours; Day 29: pre- and post-dialysis; Day 57: pre- and post-dialysis, 3, 12, 24 hours and Week 10: pre- and post-dialysis
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Millimeters of mercury
  SBP, Baseline (Day1, predose), n=45, 43 | 135.87 (20.813) | 137.00 (16.547)
  SBP, Day 1: 3 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  SBP, Day 1: 3 hours, n=44, 43 | 140.64 (18.183) | 144.05 (22.184)
  SBP, Day1: 12 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  SBP, Day1: 12 hours, n=44, 43 | 142.05 (23.150) | 143.56 (20.566)
  SBP, Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  SBP, Day 1: 24 hours, n=41, 40 | 140.24 (20.960) | 142.05 (14.822)
  SBP, Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  SBP, Day 29: pre-dialysis, n=38, 40 | 143.05 (20.351) | 148.10 (20.445)
  SBP, Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  SBP, Day 29: post dialysis, n=38, 40 | 130.97 (20.608) | 141.93 (19.038)
  SBP, Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: pre-dialysis, n=32, 36 | 142.75 (22.599) | 151.53 (19.893)
  SBP, Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: post dialysis, n=32, 36 | 135.66 (18.314) | 141.64 (20.304)
  SBP, Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: 3 hours, n=32, 36 | 140.94 (22.623) | 148.06 (20.316)
  SBP, Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: 12 hours, n=32, 36 | 130.47 (22.492) | 145.47 (18.599)
  SBP, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: 24 hours, n=32, 36 | 143.78 (17.783) | 144.83 (15.497)
  SBP, Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  SBP, Week 10: pre-dialysis, n=42, 42 | 142.71 (20.123) | 147.12 (18.285)
  SBP, Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  SBP, Week 10: post dialysis, n=41, 42 | 138.73 (19.584) | 136.74 (22.105)
  DBP, Baseline (Day1, predose), n=45, 43 | 70.00 (10.967) | 72.05 (11.307)
  DBP, Day 1: 3 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  DBP, Day 1: 3 hours, n=44, 43 | 74.91 (12.676) | 75.53 (11.701)
  DBP, Day1: 12 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  DBP, Day1: 12 hours, n=44, 43 | 77.11 (13.784) | 77.19 (12.557)
  DBP, Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  DBP, Day 1: 24 hours, n=41, 40 | 74.22 (11.010) | 76.18 (10.318)
  DBP, Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  DBP, Day 29: pre-dialysis, n=38, 40 | 71.92 (10.794) | 77.95 (12.850)
  DBP, Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  DBP, Day 29: post dialysis, n=38, 40 | 69.47 (11.272) | 73.30 (10.823)
  DBP, Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: pre-dialysis, n=32, 36 | 72.69 (9.855) | 76.69 (12.578)
  DBP, Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: post dialysis, n=32, 36 | 71.47 (10.586) | 72.56 (10.383)
  DBP, Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: 3 hours, n=32, 36 | 72.44 (13.023) | 75.72 (11.732)
  DBP, Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: 12 hours, n=32, 36 | 67.38 (10.536) | 75.94 (10.376)
  DBP, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: 24 hours, n=32, 36 | 76.44 (12.425) | 74.81 (8.756)
  DBP, Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  DBP, Week 10: pre-dialysis, n=42, 42 | 73.86 (12.479) | 75.83 (10.087)
  DBP, Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  DBP, Week 10: post dialysis, n=41, 42 | 71.05 (12.008) | 69.52 (10.341)

53. Other Pre Specified Outcome: Absolute Values for Temperature
Description: Temperature was measured in participants in a semi-supine position after 5 minutes rest. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment.
Time Frame: as for outcome 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Degrees celsius
  Baseline (Day1, predose), n=45, 43 | 36.456 (0.3708) | 36.442 (0.3692)
  Day 1: 3 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  Day 1: 3 hours, n=44, 43 | 36.427 (0.3480) | 36.374 (0.3102)
  Day1: 12 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  Day1: 12 hours, n=44, 43 | 36.470 (0.4032) | 36.507 (0.4125)
  Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  Day 1: 24 hours, n=41, 40 | 36.459 (0.3598) | 36.380 (0.3539)
  Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: pre-dialysis, n=38, 40 | 36.389 (0.3547) | 36.418 (0.3169)
  Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: post dialysis, n=38, 40 | 36.316 (0.3576) | 36.380 (0.3040)
  Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: pre-dialysis, n=32, 36 | 36.419 (0.3685) | 36.403 (0.3410)
  Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: post dialysis, n=32, 36 | 36.384 (0.3028) | 36.378 (0.2977)
  Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 3 hours, n=32, 36 | 36.422 (0.3066) | 36.497 (0.4018)
  Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 12 hours, n=32, 36 | 36.525 (0.4363) | 36.414 (0.3474)
  Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 24 hours, n=32, 36 | 36.447 (0.3360) | 36.506 (0.3014)
  Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  Week 10: pre-dialysis, n=42, 42 | 36.414 (0.3375) | 36.383 (0.2469)
  Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  Week 10: post dialysis, n=41, 42 | 36.461 (0.3767) | 36.450 (0.2625)

54. Other Pre Specified Outcome: Absolute Values for Pulse Rate
Description: Pulse rate was measured in participants in a semi-supine position after 5 minutes rest. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment.
Time Frame: Baseline (Day 1, predose) and at Day 1:3, 12, 24 hours; Day 29: pre- and post-dialysis; Day 57: pre- and post-dialysis, 3, 12, 24 hours and Week 10: pre- and post-dialysis
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 45 | 43
Beats per minute
  Baseline (Day1, predose), n=45, 43 | 72.09 (9.860) | 76.19 (11.450)
  Day 1: 3 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  Day 1: 3 hours, n=44, 43 | 72.48 (9.931) | 76.21 (10.432)
  Day1: 12 hours, n=44, 43: number analyzed (Participants) | 44 | 43
  Day1: 12 hours, n=44, 43 | 71.95 (9.101) | 72.65 (9.564)
  Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  Day 1: 24 hours, n=41, 40 | 73.37 (10.495) | 76.43 (8.388)
  Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: pre-dialysis, n=38, 40 | 72.92 (11.751) | 76.05 (8.688)
  Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: post dialysis, n=38, 40 | 74.00 (10.051) | 76.18 (11.437)
  Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: pre-dialysis, n=32, 36 | 74.59 (12.793) | 77.17 (10.997)
  Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: post dialysis, n=32, 36 | 72.63 (10.354) | 75.75 (9.927)
  Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 3 hours, n=32, 36 | 70.91 (11.360) | 75.25 (9.755)
  Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 12 hours, n=32, 36 | 70.50 (11.259) | 75.11 (9.858)
  Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 24 hours, n=32, 36 | 71.16 (10.097) | 75.36 (7.650)
  Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  Week 10: pre-dialysis, n=42, 42 | 73.07 (10.744) | 75.81 (9.823)
  Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  Week 10: post dialysis, n=41, 42 | 71.76 (10.138) | 74.55 (11.096)

55. Other Pre Specified Outcome: Change From Baseline Values for Vital Signs: SBP and DBP
Description: Vital signs including SBP and DBP were measured in participants in a semi-supine position after 5 minutes rest. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: as for outcome 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 44 | 43
Millimeters of mercury
  SBP, Day 1: 3 hours, n=44, 43 | 5.34 (20.307) | 7.05 (18.639)
  SBP, Day1: 12 hours, n=44, 43 | 6.75 (25.642) | 6.56 (17.633)
  SBP, Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  SBP, Day 1: 24 hours, n=41, 40 | 3.90 (21.846) | 6.23 (18.150)
  SBP, Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  SBP, Day 29: pre-dialysis, n=38, 40 | 8.24 (27.069) | 12.00 (25.314)
  SBP, Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  SBP, Day 29: post dialysis, n=38, 40 | -3.84 (20.676) | 5.83 (21.882)
  SBP, Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: pre-dialysis, n=32, 36 | 6.63 (25.125) | 16.03 (20.492)
  SBP, Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: post dialysis, n=32, 36 | -0.47 (22.747) | 6.14 (20.699)
  SBP, Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: 3 hours, n=32, 36 | 4.81 (22.938) | 12.56 (20.832)
  SBP, Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: 12 hours, n=32, 36 | -5.66 (25.575) | 9.97 (20.520)
  SBP, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  SBP, Day 57: 24 hours, n=32, 36 | 7.66 (21.919) | 9.33 (22.080)
  SBP, Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  SBP, Week 10: pre-dialysis, n=42, 42 | 7.36 (21.412) | 10.48 (19.261)
  SBP, Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  SBP, Week 10: post dialysis, n=41, 42 | 2.73 (19.005) | 0.10 (23.472)
  DBP, Day 1: 3 hours, n=44, 43 | 5.07 (12.617) | 3.49 (13.170)
  DBP, Day1: 12 hours, n=44, 43 | 7.27 (13.588) | 5.14 (13.105)
  DBP, Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  DBP, Day 1: 24 hours, n=41, 40 | 4.07 (13.129) | 4.18 (11.569)
  DBP, Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  DBP, Day 29: pre-dialysis, n=38, 40 | 2.63 (14.749) | 5.88 (14.650)
  DBP, Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  DBP, Day 29: post dialysis, n=38, 40 | 0.18 (13.854) | 1.23 (12.259)
  DBP, Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: pre-dialysis, n=32, 36 | 2.94 (13.457) | 5.86 (13.316)
  DBP, Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: post dialysis, n=32, 36 | 1.72 (11.277) | 1.72 (12.230)
  DBP, Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: 3 hours, n=32, 36 | 2.69 (17.087) | 4.89 (14.540)
  DBP, Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: 12 hours, n=32, 36 | -2.38 (13.760) | 5.11 (14.186)
  DBP, Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  DBP, Day 57: 24 hours, n=32, 36 | 6.69 (15.995) | 3.97 (13.729)
  DBP, Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  DBP, Week 10: pre-dialysis, n=42, 42 | 3.71 (13.328) | 3.50 (12.975)
  DBP, Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  DBP, Week 10: post dialysis, n=41, 42 | 1.00 (10.151) | -2.81 (12.934)

56. Other Pre Specified Outcome: Change From Baseline Values for Temperature
Description: Temperature was measured in participants in a semi-supine position after 5 minutes rest. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: as for outcome 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Degrees celsius
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 44 | 43
Degrees celsius
  Day 1: 3 hours, n=44, 43 | -0.027 (0.3744) | -0.067 (0.3220)
  Day1: 12 hours, n=44, 43 | 0.016 (0.4011) | 0.065 (0.3981)
  Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  Day 1: 24 hours, n=41, 40 | 0.015 (0.3712) | -0.050 (0.3359)
  Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: pre-dialysis, n=38, 40 | -0.089 (0.5451) | -0.033 (0.3731)
  Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: post dialysis, n=38, 40 | -0.163 (0.4790) | -0.070 (0.4027)
  Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: pre-dialysis, n=32, 36 | -0.003 (0.4447) | -0.028 (0.4158)
  Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: post dialysis, n=32, 36 | -0.038 (0.3774) | -0.053 (0.3247)
  Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 3 hours, n=32, 36 | 0.000 (0.4048) | 0.067 (0.4697)
  Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 12 hours, n=32, 36 | 0.103 (0.5196) | -0.017 (0.3085)
  Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 24 hours, n=32, 36 | 0.025 (0.4501) | 0.075 (0.3557)
  Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  Week 10: pre-dialysis, n=42, 42 | -0.055 (0.4840) | -0.062 (0.4328)
  Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  Week 10: post dialysis, n=41, 42 | -0.002 (0.5270) | 0.005 (0.4311)

57. Other Pre Specified Outcome: Change From Baseline Values for Pulse Rate
Description: Pulse rate was measured in participants in a semi-supine position after 5 minutes rest. Baseline (Day 1-predose) is the latest non-missing pre-dose assessment. Change from Baseline is defined as Post-dose visit value minus Baseline value.
Time Frame: as for outcome 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
Number analyzed (Participants) | 44 | 43
Beats per minute
  Day 1: 3 hours, n=44, 43 | 0.61 (7.735) | 0.02 (10.859)
  Day1: 12 hours, n=44, 43 | 0.09 (8.232) | -3.53 (12.473)
  Day 1: 24 hours, n=41, 40: number analyzed (Participants) | 41 | 40
  Day 1: 24 hours, n=41, 40 | 1.39 (10.954) | -0.35 (11.005)
  Day 29: pre-dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: pre-dialysis, n=38, 40 | 0.87 (9.393) | 0.03 (10.850)
  Day 29: post dialysis, n=38, 40: number analyzed (Participants) | 38 | 40
  Day 29: post dialysis, n=38, 40 | 1.95 (11.203) | 0.15 (12.593)
  Day 57: pre-dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: pre-dialysis, n=32, 36 | 2.50 (10.522) | 2.14 (10.805)
  Day 57: post dialysis, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: post dialysis, n=32, 36 | 0.53 (9.308) | 0.72 (12.523)
  Day 57: 3 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 3 hours, n=32, 36 | -1.19 (11.998) | 0.22 (12.547)
  Day 57: 12 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 12 hours, n=32, 36 | -1.59 (12.104) | 0.08 (10.811)
  Day 57: 24 hours, n=32, 36: number analyzed (Participants) | 32 | 36
  Day 57: 24 hours, n=32, 36 | -0.94 (11.435) | 0.33 (10.368)
  Week 10: pre-dialysis, n=42, 42: number analyzed (Participants) | 42 | 42
  Week 10: pre-dialysis, n=42, 42 | 1.33 (10.195) | -0.48 (13.457)
  Week 10: post dialysis, n=41, 42: number analyzed (Participants) | 41 | 42
  Week 10: post dialysis, n=41, 42 | -0.54 (9.344) | -1.74 (11.232)

ADVERSE EVENTS:
Time Frame: Non-SAEs were reported from start of study treatment and up to 8 weeks in treatment period and SAEs were reported from the start of the study treatment and up to 2 weeks in follow up period (Up to Week 10).
Description: Non-SAEs and SAEs were reported for Safety Population.
Arm/Group | Daprodustat | Recombinant Human Erythropoietin
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 10/45 | 5/43
Other Adverse Events (participants affected / at risk) | 10/45 | 4/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=45) | Recombinant Human Erythropoietin (N=43)
Fluid overload (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=45) | Recombinant Human Erythropoietin (N=43)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (6)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03029247/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT03029247/SAP_001.pdf